

# A PHASE 2, RANDOMIZED, OPEN-LABEL TRIAL TO EVALUATE THE SAFETY AND IMMUNOGENICITY OF A MULTIVALENT PNEUMOCOCCAL CONJUGATE VACCINE GIVEN WITH, OR SEPARATELY FROM, 13-VALENT PNEUMOCOCCAL CONJUGATE VACCINE IN HEALTHY INFANTS

**Investigational Product Number:** PF-06842433

**Investigational Product Name:** Complementary 7-valent Pneumococcal

Conjugate Vaccine

**United States (US) Investigational New** 

**Drug (IND) Number:** 

CCI

**European Clinical Trials Database** 

(EudraCT) Number:

Protocol Number: C3571002

Phase: 2

This document and accompanying materials contain confidential information belonging to Pfizer. Except as otherwise agreed to in writing, by accepting or reviewing these documents, you agree to hold this information in confidence and not copy or disclose it to others (except where required by applicable law) or use it for unauthorized purposes. In the event of any actual or suspected breach of this obligation, Pfizer must be promptly notified.

# **Document History**

| Document | Version Date | Summary of Changes and Rationale |
|---|---|---|
| Amendment 1 | 18 Feb 2020 | Title Page: Added the US IND number, which was pending at the time of protocol finalization. |
| | | Protocol Summary and Section 3:<br>Removed the consideration of sites<br>from other countries outside of the<br>United States as only US sites are<br>participating in the study. |
| | | Protocol Summary and Section 3:<br>Updated the total number of subjects<br>randomized from "approximately<br>690" to "565" due to the adequacy<br>of this study size to provide the<br>needed information to evaluate the<br>endpoints and facilitate a timely<br>readout for this descriptive study.<br>The number of subjects per arm was<br>also updated accordingly. |
| | | Section 4.2: Reworded exclusion criterion 5 to, "Prior receipt of hepatitis B vaccine at age ≥30 days" to further clarify the criterion. |
| | | Section 5.7.3: Clarified that a licensed inactivated influenza vaccine may be given to eligible study subjects during influenza season. |
| | | Section 6: Clarified that the subject's recorded demographic information will include race. |
| | | Section 8.2.1: Clarified that events consistent with normal growth and development are generally not to be considered adverse events. |
| | | Sections 9.1, 9.3.1, and 9.3.2:<br>Updated the number of subjects per arm and the probabilities of detecting AEs by frequency, |

Final Protocol Amendment 1, 18 Feb 2020

| Document | Version Date | Summary of Changes and Rationale |
|-------------------|--------------|----------------------------------|
| Original protocol | 21 Dec 2017 | Not applicable (N/A) |

This amendment incorporates all revisions to date, including amendments made at the request of the country health authorities and institutional review boards (IRBs)/ethics committee (ECs).

# **TABLE OF CONTENTS**

| LIST OF TABLES | 9 |
|---------------------------------------------------------|----|
| APPENDICES | 9 |
| PROTOCOL SUMMARY | 10 |
| SCHEDULE OF ACTIVITIES | 14 |
| 1. INTRODUCTION | 20 |
| 1.1. Indication | 20 |
| 1.2. Background and Rationale | 20 |
| 1.2.1. Pneumococcal Disease | 20 |
| 1.2.2. Vaccines to Prevent Pneumococcal Disease | 21 |
| 1.2.2.1. Pneumococcal Polysaccharide Vaccines | 21 |
| 1.2.2.2. Pneumococcal Polysaccharide Conjugate Vaccines | 21 |
| 1.2.2.3. Rationale for c7vPnC | 22 |
| 2. STUDY OBJECTIVES AND ENDPOINTS | 23 |
| 2.1. Primary Objective and Endpoints | 23 |
| 2.1.1. Primary Objective | 23 |
| 2.1.2. Primary Endpoints | 23 |
| 2.2. Secondary Objective and Endpoints | 24 |
| 2.2.1. Secondary Objective | 24 |
| 2.2.2. Secondary Endpoints | 24 |
| CCI | |
| 3. STUDY DESIGN | 25 |
| 3.1. Duration of Subject Participation | 26 |
| 3.2. Duration of Study | 26 |
| 3.3. Number of Subjects | 26 |
| 4. SUBJECT ELIGIBILITY CRITERIA | 27 |
| 4.1. Inclusion Criteria | 27 |
| 4.2. Exclusion Criteria | 27 |
| 4.3. Temporary Delay Criteria | 29 |

| 4.3.1. Criteria for Temporarily Delaying Dose Administration (Doses 1, 2, 3, and 4 and the Supplemental Dose) | 29 |
|---|---|
| 4.3.2. Criteria for Temporarily Delaying Blood Draw (Prior to Dose 3, 1 Month After Dose 3, Prior to Dose 4, and 1 Month After Dose 4 and the Supplemental Dose) | 29 |
| 4.4. Sponsor's Qualified Medical Personnel | 29 |
| 5. INVESTIGATIONAL PRODUCTS | 30 |
| 5.1. Allocation to Investigational Product | 30 |
| 5.2. Subject Compliance | 30 |
| 5.3. Investigational Product Supplies | 30 |
| 5.3.1. Dosage Form(s) and Packaging | 30 |
| 5.3.2. Preparation and Dispensing | 31 |
| 5.4. Administration. | 31 |
| 5.5. Investigational Product Storage | 32 |
| 5.6. Investigational Product Accountability | 33 |
| 5.6.1. Destruction of Investigational Product Supplies | 33 |
| 5.7. Concomitant Vaccines/Medications | 33 |
| 5.7.1. Concomitant Vaccines to Be Administered at Study Visits | 33 |
| 5.7.2. Prohibited Vaccines/Medications During the Study | 33 |
| 5.7.3. Permitted Vaccines/Medications During the Study | 34 |
| 5.7.4. Recording Prior and Concomitant Treatments | 34 |
| 6. STUDY PROCEDURES | 35 |
| 6.1. Group 1 (Coadministration) Study Procedures | 35 |
| 6.1.1. Group 1 Visit 1 (Dose 1: 2-Month Visit, Day 1) | 35 |
| 6.1.2. Group 1 Visit 2 (Dose 2: 4-Month Visit, 42 to 63 Days After Dose 1) | 36 |
| 6.1.3. Group 1 Visit 3 (Dose 3: 6-Month Visit, 42 to 63 Days After Dose 2) | 37 |
| 6.1.4. Group 1 Visit 4 (Follow-up: 7-Month Visit, 28 to 42 Days After Dose 3) | 38 |
| 6.1.5. Group 1 Visit 5 (Dose 4: 12-Month Visit, 365 to 386 Days of Age) | 39 |
| 6.1.6. Group 1 Visit 6 (Follow-up: 13-Month Visit, 28 to 42 Days After Dose 4) | 40 |
| 6.1.7. Group 1 Visit 7 (Follow-up: 18-Month Phone Contact, 168 to 196 Days After Dose 4) | 41 |
| 6.2. Group 2 (Staggered Administration) Study Procedures | 41 |

Final Protocol Amendment 1, 18 Feb 2020

| 7. ASSESSMENTS | 60 |
|---|---|
| 7.1. Safety Parameters | 60 |
| 7.1.1. Subject Electronic Diary | 60 |
| 7.1.2. Grading Scale for Prompted Events | 61 |
| 7.1.2.1. Local Reactions | 61 |
| 7.1.2.2. Systemic Event Symptoms and Fever | 62 |
| CCI | |
| 7.2. Immunogenicity | |
| 7.3. Biological Samples | 65 |
| CCI | |
| 8. ADVERSE EVENT REPORTING | 67 |
| 8.1. Requirements | 67 |
| 8.1.1. Additional Details on Recording Adverse Events on the CRF | 68 |
| 8.1.2. Eliciting Adverse Event Information | 68 |
| 8.1.3. Withdrawal From the Study Due to Adverse Events (see also the Subject Withdrawal Section) | 68 |
| 8.1.4. Time Period for Collecting AE/SAE/NDCMC Information | 68 |
| 8.1.4.1. Reporting SAEs to Pfizer Safety | 69 |
| 8.1.4.2. Recording Nonserious AEs and SAEs on the CRF | 69 |
| 8.1.5. Causality Assessment | 69 |
| 8.1.6. Sponsor's Reporting Requirements to Regulatory Authorities | 70 |
| 8.2. Definitions | 70 |
| 8.2.1. Adverse Events | 70 |
| 8.2.2. Abnormal Test Findings | 71 |
| 8.2.3. Serious Adverse Events | 71 |
| 8.2.4. Hospitalization | 72 |
| 8.3. Severity Assessment | 73 |
| 8.4. Special Situations | 74 |
| 8.4.1. Protocol-Specified Serious Adverse Events | 74 |
| 8.4.2. Potential Cases of Drug-Induced Liver Injury | 74 |
| 8.4.3. Exposure to the Investigational Product During Pregnancy or Breastfeeding, and Occupational Exposure | 76 |
| 8.4.3.1. Exposure During Pregnancy | 76 |

| 8.4.3.2. Exposure During Breastfeeding | 77 |
|---|---|
| 8.4.3.3. Occupational Exposure | 77 |
| 8.4.4. Medication Errors and Lack of Efficacy | 77 |
| 8.4.4.1. Medication Errors | 78 |
| 8.4.4.2. Lack of Efficacy | 78 |
| 8.5. Medical Device Complaint Reporting Requirements | 79 |
| 9. DATA ANALYSIS/STATISTICAL METHODS | 79 |
| 9.1. Sample Size Determination | 79 |
| 9.2. Analysis Populations | 79 |
| 9.3. Immunogenicity Analysis | 81 |
| 9.3.1. Analyses of Secondary CCl Endpoints | 81 |
| CCI | |
| 9.4. Safety Analysis | 83 |
| CCI | |
| 10. QUALITY CONTROL AND QUALITY ASSURANCE | 84 |
| 11. DATA HANDLING AND RECORD KEEPING | 85 |
| 11.1. Case Report Forms/Electronic Data Record | 85 |
| 11.2. Record Retention | 86 |
| 12. ETHICS | 86 |
| 12.1. Institutional Review Board/Ethics Committee | 86 |
| 12.2. Ethical Conduct of the Study | 86 |
| 12.3. Subject Information and Consent | 87 |
| 12.4. Reporting of Safety Issues and Serious Breaches of the Protocol or ICH | |
| GCP | |
| 13. DEFINITION OF END OF TRIAL | |
| 13.1. End of Trial in All Participating Countries | 88 |
| 14. SPONSOR DISCONTINUATION CRITERIA | |
| 15. PUBLICATION OF STUDY RESULTS | 88 |
| 15.1. Communication of Results by Pfizer | 88 |
| 15.2. Publications by Investigators | 89 |
| 16. REFERENCES | 91 |

# 

#### PROTOCOL SUMMARY

#### **Background and Rationale**

Streptococcus pneumoniae are gram-positive encapsulated cocci that are a leading cause of bacteremia, bacterial meningitis, pneumonia, and acute otitis media (AOM) and continue to be a major global public health concern. Serious pneumococcal disease may occur at any age; however, children <5 years and adults ≥65 years of age are at particularly increased risk. Individuals with certain comorbidities and immunocompromising conditions are also at risk, especially persons with chronic heart, lung, liver, and renal disease, as well as those who are functionally asplenic. AOM carries the risk of complications such as tympanostomy tube placement, hearing loss, mastoiditis, and meningitis as well as being a significant burden on the healthcare system. S pneumoniae remains an important cause of serious disease in the United States and worldwide.

The polysaccharide capsule has been identified as an important virulence factor for this pathogen. While more than 95 pneumococcal serotypes, differentiated by their capsular polysaccharide composition, have been identified, serious disease is generally caused by a smaller subset of serotypes. Pneumococcal disease can be prevented with polysaccharidebased vaccines that induce antibody responses with functional (opsonophagocytic) activity and target the capsular serotypes responsible for disease. Pneumococcal vaccines containing free polysaccharides, such as the licensed 23-valent pneumococcal polysaccharide vaccine (PPSV23), are poorly immunogenic in immunocompromised populations, older adults, and children less than 2 years of age, and are not recommended in this younger age group. This led to development of pneumococcal conjugate vaccines, which contain capsular polysaccharides covalently linked to a protein carrier, and which induce protective immune responses in young children and older adults, as well as populations with high-risk conditions. Prevnar® (7-valent pneumococcal conjugate vaccine), which was licensed in the United States in 2000, and Prevnar 13® (13-valent pneumococcal conjugate vaccine), which was licensed in the United States in 2010, are pneumococcal conjugate vaccines containing 7 and 13 pneumococcal capsular polysaccharides, respectively, that are each covalently linked to a nontoxic variant of diphtheria toxin, cross-reactive material ( $CRM_{197}$ ). These vaccines targeted serotypes that caused the majority of pneumococcal disease in infants and older adults at the time of their introduction. They have demonstrated efficacy/effectiveness against vaccine-type (VT) invasive pneumococcal disease (IPD) such as bacteremia and meningitis, as well as AOM, and community-acquired pneumonia (CAP). Additionally, they have been found to reduce nasopharyngeal carriage and transmission, resulting in beneficial indirect effects.

Pfizer is developing a new complementary 7-valent pneumococcal conjugate vaccine (c7vPnC) candidate to expand protection against pneumococcal disease beyond that covered by current pneumococcal vaccines in children and adults. c7vPnC contains pneumococcal conjugates of 7 different serotypes (8, 10A, 11A, 12F, 15B, 22F, and 33F). c7vPnC contains the same conjugate carrier protein and excipients and uses the same platform as Prevnar 13. A meta-analysis of serotypes causing IPD in children <5 years of age in regions of the world that have introduced higher-valent pneumococcal conjugate vaccines (such as Prevnar 13) showed that, overall, these 7 serotypes accounted for approximately 70% of disease not due



The purpose of this Phase 2 study is to describe the safety and immunogenicity of c7vPnC coadministered with Prevnar 13 in infants at 2, 4, 6, and 12 months of age or given 1 month after Prevnar 13 at 3, 5, 7, and 13 months of age.

Safety and immunogenicity data from this study will inform further clinical development of c7vPnC in pediatric populations.

Additional information for this compound may be found in the single reference safety document (SRSD), which for this study is the c7vPnC investigator's brochure (IB). The SRSD for Prevnar 13 is the US package insert (USPI).

#### **Study Design**

This is a Phase 2, multicenter, randomized, active-controlled, open-label study with a 3-arm parallel design. It is planned to be conducted at investigator sites in the United States. A total of 565 infants aged  $\geq$ 42 to  $\leq$ 98 days will be randomized (1:1:1) to receive a vaccine series with:

- c7vPnC coadministered with Prevnar 13 (Group 1 coadministration);
- c7vPnC given 1 month after Prevnar 13 (Group 2 staggered administration); or
- Prevnar 13 alone as the active control group (Group 3 control with Supplemental Dose). A single dose of c7vPnC will be administered after the Prevnar 13 series is completed in this group.

In all groups, Prevnar 13 will be administered at 2, 4, 6, and 12 months of age. c7vPnC will be administered at 2, 4, 6, and 12 months of age in Group 1; at 3, 5, 7, and 13 months of age in Group 2; and at 13 months of age in Group 3. **Note:** In this document, and related study documents, vaccine (investigational product) Doses 1, 2, 3, and 4 specifically refer to the doses of c7vPnC administered in Groups 1 and 2, or the doses of Prevnar 13 administered in the control group (Group 3). The dose of c7vPnC in Group 3 will be referred to as the Supplemental Dose.

Vaccine containing diphtheria, tetanus, and acellular pertussis antigens will be administered at 2, 4, and 6 months of age. This is part of routine standard of care in the United States,

Other routine pediatric vaccines may be administered in this study, with or without certain restrictions. Local

reactions (redness, swelling, and pain) at the injection site and systemic events (fever, decreased appetite, drowsiness/increased sleep, and irritability) will be prompted for and collected by an electronic diary (e-diary; device or application) from Day 1 to Day 7 following Doses 1 to 4 and the Supplemental Dose. Use of antipyretic/pain medications from Day 1 to Day 7 following vaccination will also be collected by an e-diary. Adverse events (AEs) will be collected from the time of informed consent to 1 month after Dose 3 and from Dose 4 to 1 month after Dose 4 or 1 month after the Supplemental Dose in Group 3. Serious adverse events (SAEs) and newly diagnosed chronic medical conditions (NDCMCs) will be collected from the time of informed consent through 6 months after Dose 4 or the Supplemental Dose. Blood will be drawn for immunogenicity assessments 1 month after Dose 3, prior to receipt of Dose 4, and 1 month after Dose 4 CCI.

In Group 2, blood will also be collected prior to Dose 3. See Section 3, Table 1, for an overview of the vaccinations and blood draws in the study.



#### **Primary Objective and Endpoints**

#### **Primary Objective**

• To describe the safety profile of c7vPnC in healthy infants.

#### **Primary Endpoints**

- Proportions of subjects reporting prompted local reactions (redness, swelling, and pain at the injection site) within 7 days of each dose.
- Proportions of subjects reporting prompted systemic events (fever, decreased appetite, drowsiness/increased sleep, and irritability) within 7 days of each dose.
- Proportions of subjects reporting AEs from Dose 1 to 1 month following Dose 3 and from Dose 4 to 1 month following Dose 4/Supplemental Dose.
- Proportions of subjects reporting SAEs and NDCMCs from Dose 1 to 6 months following Dose 4/Supplemental Dose.

#### **Secondary Objective and Endpoints**

#### **Secondary Objective**

• To describe the immunogenicity of c7vPnC in healthy infants.

#### **Secondary Endpoints**

• Pneumococcal serotype-specific immunoglobulin G (IgG) concentrations 1 month after Dose 3.

• Pneumococcal serotype-specific IgG concentrations 1 month after Dose 4.



#### **Statistical Methods**

An analysis of safety and immunogenicity data will be conducted when data are available as described in Section 9 according to the statistical analysis plan (SAP). All analyses will be descriptive. No hypothesis tests between vaccine groups are planned; therefore, no power calculations for comparison of vaccine groups are included.

#### **SCHEDULE OF ACTIVITIES**

The schedule of activities table provides an overview of the protocol visits and procedures. Refer to the Study Procedures and Assessments sections of the protocol for detailed information on each procedure and assessment required for compliance with the protocol.

The investigator may schedule visits (unplanned visits) in addition to those listed on the schedule of activities table, in order to conduct evaluations or assessments required to protect the well-being of the subject.

**Group 1 – Coadministration** 

| Visit Number | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
|---|---|---|---|---|---|---|---|
| Visit Description | Dose 1<br>2-Month Visit | Dose 2<br>4-Month Visit | Dose 3<br>6-Month Visit | Follow-up<br>7-Month Visit | Dose 4<br>12-Month Visit | Follow-up<br>13-Month Visit | Follow-up Phone<br>Call<br>18-Month Phone<br>Contact |
| Visit Window (Days) | Day 1 | 42 to 63 Days<br>After Dose 1 | 42 to 63 Days<br>After Dose 2 | 28 to 42 Days<br>After Dose 3 | 365 to 386 Days<br>of Age | 28 to 42 Days<br>After Dose 4 | 168 to 196 Days<br>After Dose 4 |
| Obtain informed consent | X | | | | | | |
| Record demography | X | | | | | | |
| Obtain medical history data | X | | | | | | |
| Perform physical examination | X | | | | | | |
| Obtain prevaccination rectal temperature | X | X | X | | X | | |
| Record prior and interim vaccinations | X | X | X | X | X | X | |
| Review inclusion and exclusion criteria | X | | | | | | |
| Review temporary delay criteria | X | X | X | X | X | X | |
| Review continued eligibility | | X | X | X | X | X | |
| Assign subject number and randomization number | X | | | | | | |
| Obtain blood sample (~5 mL) | | | | X | Xa | X | |
| Administer c7vPnC (in left thigh) and Prevnar 13 (in right thigh) | X | X | X | | X | | |
| Administer DTaP-containing vaccine (at site other than left leg) <sup>b</sup> | X | X | X | | | | |
| Administer other permitted concomitant vaccines (at site other than left leg) <sup>b</sup> | X | X | X | | X | | |
| Assess and record acute reactions for at least 30 minutes after vaccine administration | X | X | X | | X | | |

| Visit Number | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
|---|---|---|---|---|---|---|---|
| Visit Description | Dose 1<br>2-Month Visit | Dose 2<br>4-Month Visit | Dose 3<br>6-Month Visit | Follow-up<br>7-Month Visit | Dose 4<br>12-Month Visit | Follow-up<br>13-Month Visit | Follow-up Phone<br>Call<br>18-Month Phone<br>Contact |
| Visit Window (Days) | Day 1 | 42 to 63 Days | 42 to 63 Days | 28 to 42 Days | 365 to 386 Days | 28 to 42 Days | 168 to 196 Days |
| | | After Dose 1 | After Dose 2 | After Dose 3 | of Age | After Dose 4 | After Dose 4 |
| Provide subject's legally acceptable representative with an e-diary (device or application), thermometer, and measuring device and instruct how to collect prompted local reactions, systemic events, and antipyretic/pain medication use until Day 7 <sup>c</sup> | X | | | | X | | |
| Review e-diary events d,e | | X | X | X | | X | |
| Collect e-diary (if device provided) | | | | X | | X | |
| Record and report adverse events | X | | | X | X | X | |
| Record and report serious adverse events and newly diagnosed chronic medical conditions fig. | X | | | | | | X |

Abbreviations: DTaP = diphtheria, tetanus, and acellular pertussis; e-diary = electronic diary; NDCMC = newly diagnosed chronic medical condition.

- a. Blood sample will be collected prior to vaccination.
- b. The subject may receive vaccines with inactivated poliovirus, hepatitis B, or *Haemophilus influenzae* type b (either separately or in the diphtheria, tetanus, and pertussis combination vaccine) at 2, 4, and 6 months of age. Measles, mumps, and rubella (MMR) vaccination may be administered concomitantly at 12 months of age or according to the permitted treatment windows in Section 5.7.3. Rotavirus vaccine may be administered orally at any time.
- c. The subject's legally acceptable representative will record prompted local reactions and systemic events in an e-diary for the 7 days following each dose of c7vPnC. The subject's legally acceptable representative will be instructed to contact the study staff if the subject experiences redness or swelling >14 caliper units, severe pain at the injection site, or a fever >104.0°F (>40.0°C), or has an emergency room visit or hospitalization.
- d. Designated site staff will review e-diary data online at frequent intervals (daily is optimal) for the 7 days following each dose of c7vPnC to evaluate subject compliance and reported events as part of the ongoing safety review.
- f. Record concomitant medications used to treat SAEs and NDCMCs as described in Section 5.7.4.
- g. A newly diagnosed chronic medical condition is defined as a disease or medical condition, not previously identified, that is expected to be persistent or otherwise long-lasting in its effects.

# **Group 2 – Staggered Administration**

| Visit Number | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit Description | Prevnar<br>13<br>2-Month<br>Visit | c7vPnC<br>Dose 1<br>3-Month<br>Visit | Prevnar<br>13<br>4-Month<br>Visit | c7vPnC<br>Dose 2<br>5-Month<br>Visit | Prevnar<br>13<br>6-Month<br>Visit | c7vPnC<br>Dose 3<br>7-Month<br>Visit | Follow-up<br>8-Month<br>Visit | 13<br>12-<br>Month<br>Visit | c7vPnC<br>Dose 4<br>13-Month<br>Visit | Visit | up Phone<br>Call<br>19-Month<br>Phone<br>Contact |
| Visit Window (Days) | Day 1 | 21 to 35<br>Days<br>After<br>Prevnar<br>13 at<br>Visit 1 | 42 to 63<br>Days<br>After<br>Prevnar<br>13 at<br>Visit 1 | 21 to 35<br>Days<br>After<br>Prevnar<br>13 at<br>Visit 3 | 42 to 63 Days After Prevnar 13 at Visit 3 | 21 to 35<br>Days<br>After<br>Prevnar<br>13 at<br>Visit 5 | 28 to 42<br>Days<br>After<br>Dose 3 | 365 to<br>386 Days<br>of Age | 21 to 35<br>Days<br>After<br>Prevnar<br>13 at<br>Visit 8 | 28 to 42<br>Days<br>After<br>Dose 4 | 168 to<br>196 Days<br>After<br>Dose 4 |
| Obtain informed consent | X | | | | | | | | | | |
| Record demography | X | | | | | | | | | | |
| Obtain medical history data | X | | | | | | | | | | |
| Perform physical examination | X | | | | | | | | | | |
| Obtain prevaccination rectal temperature | | X | | X | | X | | | X | | |
| Record prior and interim vaccinations | X | X | X | X | X | X | X | X | X | X | |
| Review inclusion and exclusion criteria | X | | | | | | | | | | |
| Review temporary delay criteria | | X | | X | | X | X | | X | X | |
| Review continued eligibility | | X | X | X | X | X | X | X | X | X | |
| Assign subject number and randomization number | X | | | | | | | | | | |
| Obtain blood sample (~5 mL) | | | | | | Xª | X | | Xª | X | |
| Administer Prevnar 13 (in right thigh) | X | | X | | X | | | X | | | |
| Administer c7vPnC (in left thigh) | | X | | X | | X | | | X | | |
| Administer DTaP-containing vaccine (at site other than left leg) <sup>b</sup> | X | | X | | X | | | | | | |
| Administer other permitted concomitant vaccines (at site other than left leg) <sup>b</sup> | X | | X | | X | | | X | | | |
| Assess and record acute reactions for at least 30 minutes after vaccine administration | | X | | X | | X | | | X | | |
| Provide subject's legally acceptable representative with an e-diary (device or application), thermometer, and measuring device and instruct how to collect prompted local reactions, systemic events, and antipyretic/pain medication use until Day 7° | | X | | | | | | | X | | |

| Visit Number | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit Description | Prevnar | c7vPnC | Prevnar | c7vPnC | Prevnar | c7vPnC | Follow-up | Prevnar | c7vPnC | Follow-up | Follow- |
| | 13 | Dose 1 | 13 | Dose 2 | 13 | Dose 3 | 8-Month | 13 | Dose 4 | 14-Month | up Phone |
| | 2-Month | 3-Month | 4-Month | 5-Month | 6-Month | 7-Month | Visit | 12- | 13-Month | Visit | Call |
| | Visit | Visit | Visit | Visit | Visit | Visit | | Month | Visit | | 19-Month |
| | | | | | | | | Visit | | | Phone |
| | | | | | | | | | | | Contact |
| Visit Window (Days) | Day 1 | 21 to 35 | 42 to 63 | 21 to 35 | 42 to 63 | 21 to 35 | 28 to 42 | 365 to | 21 to 35 | 28 to 42 | 168 to |
| | | Days | Days | Days | Days | Days | Days | <b>386 Days</b> | Days | Days | <b>196 Days</b> |
| | | After | After | After | After | After | After | of Age | After | After | After |
| | | Prevnar | Prevnar | Prevnar | Prevnar | Prevnar | Dose 3 | | Prevnar | Dose 4 | Dose 4 |
| | | 13 at | 13 at | 13 at | 13 at | 13 at | | | 13 at | | |
| | | Visit 1 | Visit 1 | Visit 3 | Visit 3 | Visit 5 | | | Visit 8 | | |
| Review e-diary events <sup>d,e</sup> | | | X | | X | | X | | | X | |
| Collect e-diary (if device provided) | | | | | | | X | | | X | |
| Record and report adverse events | X | | | | | | X | | X | X | |
| Record and report serious adverse events and newly diagnosed chronic medical conditions <sup>f,g</sup> | X- | | | | | | | | | | ·-X |

Abbreviations: DTaP = diphtheria, tetanus, and acellular pertussis; e-diary = electronic diary; NDCMC = newly diagnosed chronic medical condition.

- a. Blood sample will be collected prior to vaccination.
- b. The subject may receive vaccines with inactivated poliovirus, hepatitis B, or *Haemophilus influenzae* type b (either separately or in the diphtheria, tetanus, and pertussis combination vaccine) at 2, 4, and 6 months of age. Measles, mumps, and rubella (MMR) vaccination may be administered concomitantly at 12 months of age or according to the permitted treatment windows in Section 5.7.3. Rotavirus vaccine may be administered orally at any time.
- c. The subject's legally acceptable representative will record prompted local reactions and systemic events in an e-diary for the 7 days following each dose of c7vPnC. The subject's legally acceptable representative will be instructed to contact the study staff if the subject experiences redness or swelling >14 caliper units, severe pain at the injection site, or a fever >104.0°F (>40.0°C), or has an emergency room visit or hospitalization.
- d. Designated site staff will review e-diary data online at frequent intervals (daily is optimal) for the 7 days following each dose of c7vPnC to evaluate subject compliance and reported events as part of the ongoing safety review.
- f. Record concomitant medications used to treat SAEs and NDCMCs as described in Section 5.7.4.
- g. A newly diagnosed chronic medical condition is defined as a disease or medical condition, not previously identified, that is expected to be persistent or otherwise long-lasting in its effects.

# $Group\ 3-Control\ Group\ With\ Supplemental\ Dose$

| Visit Number | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 |
|---|---|---|---|---|---|---|---|---|
| Visit Description | Dose 1<br>2-Month Visit | Dose 2<br>4-Month Visit | Dose 3<br>6-Month Visit | Follow-up<br>7-Month Visit | Dose 4<br>12-Month Visit | Follow-up and<br>Supplemental<br>Dose<br>13-Month Visit | Follow-up of<br>Supplemental<br>Dose<br>14-Month Visit | Follow-up<br>Phone Call<br>19-Month<br>Phone Contact |
| Visit Window (Days) | Day 1 | 42 to 63 Days<br>After Dose 1 | 42 to 63 Days<br>After Dose 2 | 28 to 42 Days<br>After Dose 3 | 365 to 386<br>Days of Age | 28 to 42 Days<br>After Dose 4 | 28 to 42 Days<br>After<br>Supplemental<br>Dose | 168 to 196<br>Days After<br>Supplemental<br>Dose |
| Obtain informed consent | X | | | | | | | |
| Record demography | X | | | | | | | |
| Obtain medical history data | X | | | | | | | |
| Perform physical examination | X | | | | | | | |
| Obtain prevaccination rectal temperature | X | X | X | | X | X | | |
| Record prior and interim vaccinations | X | X | X | X | X | X | X | |
| Review inclusion and exclusion criteria | X | | | | | | | |
| Review temporary delay criteria | X | X | X | X | X | X | X | |
| Review continued eligibility | | X | X | X | X | X | X | |
| Assign subject number and randomization number | X | | | | | | | |
| Obtain blood sample (~5 mL) | | | | X | Xa | Xa | CCI | |
| Administer Prevnar 13 (in left thigh) | X | X | X | | X | | | |
| Administer DTaP-containing vaccine (at site other than left leg) <sup>b</sup> | X | X | X | | | | | |
| Administer other permitted concomitant vaccines (at site other than left leg) <sup>b</sup> | X | X | X | | X | | | |
| Administer c7vPnC (in left thigh) | | | | | | X | | |
| Assess and record acute reactions for at least 30 minutes after vaccine administration | X | X | X | | X | X | | |

| Visit Number | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 |
|---|---|---|---|---|---|---|---|---|
| Visit Description | Dose 1<br>2-Month Visit | Dose 2<br>4-Month Visit | Dose 3<br>6-Month Visit | Follow-up<br>7-Month Visit | Dose 4<br>12-Month Visit | Dose | Follow-up of<br>Supplemental<br>Dose<br>14-Month Visit | Follow-up<br>Phone Call<br>19-Month<br>Phone Contact |
| Visit Window (Days) | Day 1 | 42 to 63 Days<br>After Dose 1 | 42 to 63 Days<br>After Dose 2 | 28 to 42 Days<br>After Dose 3 | 365 to 386<br>Days of Age | 28 to 42 Days<br>After Dose 4 | 28 to 42 Days<br>After<br>Supplemental<br>Dose | 168 to 196<br>Days After<br>Supplemental<br>Dose |
| Provide subject's legally acceptable representative with an e-diary (device or application), thermometer, and measuring device and instruct how to collect prompted local reactions, systemic events, and antipyretic/pain medication use until Day 7° | X | | | | X | | 2000 | 2030 |
| Review e-diary events <sup>d</sup> | | X | X | X | | X | X | |
| Collect e-diary (if device provided) | | | | X | | | X | |
| Record and report adverse events | X | | | X | X | | X | |
| Record and report serious adverse events<br>and newly diagnosed chronic medical<br>conditions <sup>e,f</sup> | X | | | · | | | | X |

Abbreviations: DTaP = diphtheria, tetanus, and acellular pertussis; e-diary = electronic diary; NDCMC = newly diagnosed chronic medical condition.

- a. Blood sample will be collected prior to vaccination.
- b. The subject may receive vaccines with inactivated poliovirus, hepatitis B, or *Haemophilus influenzae* type b (either separately or in the diphtheria, tetanus, and pertussis combination vaccine) at 2, 4, and 6 months of age. Measles, mumps, and rubella (MMR) vaccination may be administered concomitantly at 12 months of age or according to the permitted treatment windows in Section 5.7.3. Rotavirus vaccine may be administered orally at any time.
- c. The subject's legally acceptable representative will record prompted local reactions and systemic events in an e-diary for the 7 days following each dose of Prevnar 13 and c7vPnC Supplemental Dose. For the c7vPnC Supplemental Dose only, the subject's legally acceptable representative will be instructed to contact the study staff if the subject experiences redness or swelling >14 caliper units, severe pain at the injection site, or a fever >104.0°F (>40.0°C), or has an emergency room visit or hospitalization.
- d. Designated site staff will review e-diary data online at frequent intervals (daily is optimal) for the 7 days following each dose of Prevnar 13 and c7vPnC Supplemental Dose to evaluate subject compliance and reported events as part of the ongoing safety review.
- e. Record concomitant medications used to treat SAEs and NDCMCs as described in Section 5.7.4.
- f. A newly diagnosed chronic medical condition is defined as a disease or medical condition, not previously identified, that is expected to be persistent or otherwise long-lasting in its effects.

#### 1. INTRODUCTION

#### 1.1. Indication

Complementary 7-valent pneumococcal conjugate vaccine (c7vPnC) is being developed for:

• Active immunization to prevent disease caused by the Streptococcus pneumoniae serotypes in the vaccine.

#### 1.2. Background and Rationale

#### 1.2.1. Pneumococcal Disease

S pneumoniae are gram-positive encapsulated cocci that are a leading cause of bacteremia, bacterial meningitis, pneumonia, and acute otitis media (AOM) and continue to be a major global public health concern. 1,2,3 Serious pneumococcal disease may occur at any age; however, children <5 years and adults ≥65 years of age are at particularly increased risk. Individuals with certain comorbidities and immunocompromising conditions are also at risk, especially persons with chronic heart, lung, liver, and renal disease, as well as those who are functionally asplenic. The global burden of pneumococcal disease has been substantially impacted by pneumococcal conjugate vaccines. S pneumoniae caused an estimated 14.5 million cases of serious disease and 826,000 deaths annually in children <5 years of age prior to introduction of pneumococcal conjugate vaccines. A recent estimate suggested that in 2015, several years following introduction of pneumococcal conjugate vaccines into the national infant immunization programs of more than 100 countries, the global disease burden had declined, but S pneumoniae still accounted for 2.6 million cases of severe pneumococcal disease, 332,000 deaths in children <5 years of age, and 11% of deaths in children between the ages of 1 and 5 years. 5

The overall invasive pneumococcal disease (IPD) burden was estimated in 2014 to have decreased approximately 90% in the population <5 years of age in the United States since the introduction of pneumococcal conjugate vaccines.<sup>6</sup> Even after the introduction of Prevnar 13<sup>®</sup> (13-valent pneumococcal conjugate vaccine), a significant proportion of IPD cases in persons <18 years of age is associated with hospitalization (71%), with a case fatality rate of 3%. This is due to the decrease in disease due to the serotypes in Prevnar® (7-valent pneumococcal conjugate vaccine) and Prevnar 13; however, disease due to serotypes not covered by those vaccines remains, and causes significant morbidity and mortality. Pediatric surveillance studies conducted between 2007 and 2013 in 8 US children's hospitals, and between 1997 and 2010 in a referral center in Utah, found case fatality rates of 10% and 13% with pneumococcal meningitis, respectively. These studies also found that between 52% and 63% of children surviving pneumococcal meningitis experience neurologic sequelae.<sup>8,9</sup> Surveillance studies conducted in 2010-2012 by the Centers for Disease Control and Prevention (CDC) found that S pneumoniae remains among the most common pathogens identified in community-acquired pneumonia (CAP) requiring hospitalization in the United States in both children and adults. <sup>10,11</sup> These data suggest that S pneumoniae remains an important cause of serious disease in the United States and worldwide.

AOM is a common childhood illness, with the 2011 visit rates of 0.82 and 0.81 visits for AOM/child-year in children <2 years of age and 2 to 6 years of age, respectively, and represents a significant medical burden. While AOM is generally not considered a serious disease, it does carry the risk of more serious complications. These complications can range from the development of chronic or recurrent otitis media necessitating surgical intervention (tympanostomy tube placement), and accompanied by hearing losses with potential developmental and language delays, to invasive extension leading to mastoiditis and meningitis.

Although the introduction of pneumococcal conjugate vaccines into the US and other national infant immunization programs has brought about substantial reductions in the various manifestations of pneumococcal disease in pediatric (and to some extent adult) populations, a substantial burden of pneumococcal disease remains.

#### 1.2.2. Vaccines to Prevent Pneumococcal Disease

The polysaccharide capsule has been identified as an important virulence factor for this pathogen. While more than 95 pneumococcal serotypes, differentiated by their capsular polysaccharide composition, have been identified, only a subset of serotypes are more commonly associated with severe disease. <sup>13,14</sup> Anticapsular antibodies directed against the specific serotype bind to the capsule and promote complement-mediated opsonophagocytic killing and clearance of the organism. <sup>15</sup> Pneumococcal disease can be prevented with polysaccharide-based vaccines that induce antibody responses with functional (opsonophagocytic) activity and target the capsular serotypes responsible for disease. <sup>16</sup>

#### 1.2.2.1. Pneumococcal Polysaccharide Vaccines

Vaccines containing free polysaccharides have been licensed since the 1970s. One such vaccine, 23-valent pneumococcal polysaccharide vaccine (PPSV23), has been licensed in the United States since 1983.<sup>17,18</sup> PPSV23 contains capsular polysaccharides for 23 serotypes (1, 2, 3, 4, 5, 6B, 7F, 8, 9N, 9V, 10A, 11A, 12F, 14, 15B, 17F, 18C, 19F, 19A, 20, 22F, 23F, and 33F). Pneumococcal vaccines containing free polysaccharides such as PPSV23 elicit a T-cell–independent immune response. Unconjugated polysaccharide vaccines do not induce robust responses in certain populations (eg, immunocompromised persons, children <2 years of age, and adults ≥65 years of age), nor do they generate immunologic memory, so that their protective effect wanes over 2 to 5 years.<sup>4,18,19,20</sup> Moreover, their ability to prevent nonbacteremic pneumonia, CAP, and AOM is limited or lacking.<sup>16,20,21,22,23</sup> In addition, polysaccharide vaccines do not reduce vaccine-type (VT) nasopharyngeal carriage, which is important for herd immunity.<sup>23</sup> PPSV23 is not recommended for children <2 years of age and is only recommended in children >2 years of age who are at high risk for IPD to provide some degree of protection from disease caused by serotypes not covered by existing pneumococcal conjugate vaccines.<sup>16</sup>

#### 1.2.2.2. Pneumococcal Polysaccharide Conjugate Vaccines

Pneumococcal conjugate vaccines contain polysaccharides that are covalently linked (conjugated) to an immunogenic protein. This modification results in T-cell-dependent immune responses, which have been shown to be protective in young children, older adults,

and populations with high-risk conditions. <sup>19,24</sup> Prevnar was the first pneumococcal conjugate vaccine to be licensed (2000) and was indicated for prevention of pneumococcal disease in infants and young children on the basis of efficacy studies. Prevnar contained capsular polysaccharide conjugates for 7 pneumococcal serotypes (4, 6B, 9V, 14, 18C, 19F, and 23F), each covalently linked to cross-reactive material 197 (CRM<sub>197</sub>), a nontoxic variant of diphtheria toxin. These 7 serotypes were responsible for approximately 80% to 90% of IPD in children <5 years of age in the United States and approximately 60% to 80% of IPD in the same age group in Europe at that time (1998-2000). <sup>25,26,27,28,29</sup> These serotypes also accounted for a high proportion of antibiotic-resistant strains. <sup>30</sup> Prevnar demonstrated efficacy against VT IPD, pneumonia, and AOM in large randomized, controlled efficacy studies in infants. <sup>31,32</sup> The Prevnar components contained in a related pneumococcal conjugate vaccine also were demonstrated to be efficacious against clinically/radiographically defined pneumonia. <sup>33,34,35,36</sup> Following introduction of Prevnar, reduction of nasopharyngeal carriage and transmission has resulted in indirect herd effects, with a 92% reduction of IPD due to Prevnar serotypes in older adults ≥65 years of age. <sup>37</sup>

Prevnar 13 was developed to expand serotype coverage and was licensed in the United States in 2010. Prevnar 13 includes the same *S pneumoniae* serotypes as Prevnar and an additional 6 polysaccharide conjugates for serotypes 1, 3, 5, 6A, 7F, and 19A.<sup>24,28,38</sup> The vaccine was licensed for use in infants and young children based on comparisons of serotype-specific serum immunoglobulin G (IgG) concentrations to Prevnar, with supportive data to demonstrate the functional activity of the immune responses. Prevnar 13 was later licensed in adults based on demonstration of efficacy against VT CAP in adults 65 years of age and older.<sup>39</sup> Prevnar 13 has replaced Prevnar and is licensed in the United States and many other countries, with national recommendations for use in children and older adults.<sup>40,41,42,43</sup> It has also been prequalified by the World Health Organization (WHO) for use in national infant immunization programs in lower- and middle-income countries.<sup>44,45</sup> Surveillance data from several countries following introduction of Prevnar 13 into the routine infant immunization program have demonstrated vaccine effectiveness against VT IPD in the vaccinated population.<sup>46,47,48</sup>

#### 1.2.2.3. Rationale for c7vPnC

c7vPnC is being developed to augment current pneumococcal coverage in children and adults. c7vPnC contains pneumococcal conjugates of 7 different serotypes (8, 10A, 11A, 12F, 15B, 22F, and 33F) individually conjugated to CRM<sub>197</sub>. c7vPnC uses the same platform and contains the same excipients as Prevnar and Prevnar 13. These 7 additional serotypes were selected based on their relative prevalence as a cause of IPD, their generalized geographic distribution, and other factors that would support inclusion, such as the presence of antibiotic resistance and greater disease severity (eg, meningitis, mortality). 49,50,51,52,53,54,55,56,57,58,59,60 These 7 serotypes have a long-standing association with serious pneumococcal disease. The incidence of IPD due to these 7 serotypes in children <5 years of age has remained relatively stable or slightly increased over the past several years, and these serotypes cause a significant amount of IPD in children. 61,62,63,64,65,66,67 A meta-analysis of serotypes causing IPD in children <5 years of age in regions of the world that have introduced higher-valent pneumococcal conjugate vaccines (such as Prevnar 13)

showed that, overall, these 7 serotypes accounted for approximately 70% of disease not due to the Prevnar 13 vaccine types.<sup>63</sup> Additional epidemiology data for the 7 serotypes and the preclinical program are described in the c7vPnC investigator's brochure (IB).



The purpose of this study is to assess the safety and immunogenicity of c7vPnC in infants, and to generate a safety and immunogenicity data set with c7vPnC to support and inform the design of the Phase 3 clinical development program. The targeted age of the population for this study, infants 2 months of age, has been selected as this is the indicated and recommended age of Prevnar 13 immunization in infants. Subjects will receive a 4-dose series of: c7vPnC coadministered with Prevnar 13 in Group 1; c7vPnC administered 1 month after Prevnar 13 in Group 2; or Prevnar 13 administered alone in Group 3 (control group).



Additional information for this compound may be found in the single reference safety document (SRSD), which for this study is the c7vPnC IB. The SRSD for the Prevnar 13 control vaccine is the US package insert (USPI).

#### 2. STUDY OBJECTIVES AND ENDPOINTS

#### 2.1. Primary Objective and Endpoints

#### 2.1.1. Primary Objective

• To describe the safety profile of c7vPnC in healthy infants.

#### 2.1.2. Primary Endpoints

- Proportions of subjects reporting prompted local reactions (redness, swelling, and pain at the injection site) within 7 days of each dose.
- Proportions of subjects reporting prompted systemic events (fever, decreased appetite, drowsiness/increased sleep, and irritability) within 7 days of each dose.
- Proportions of subjects reporting adverse events (AEs) from Dose 1 to 1 month following Dose 3 and from Dose 4 to 1 month following Dose 4/Supplemental Dose.

• Proportions of subjects reporting serious adverse events (SAEs) and newly diagnosed chronic medical conditions (NDCMCs) from Dose 1 to 6 months following Dose 4/Supplemental Dose.

# 2.2. Secondary Objective and Endpoints

#### 2.2.1. Secondary Objective

• To describe the immunogenicity of c7vPnC in healthy infants.

## 2.2.2. Secondary Endpoints

- Pneumococcal serotype-specific IgG concentrations 1 month after Dose 3.
- Pneumococcal serotype-specific IgG concentrations 1 month after Dose 4.



#### 3. STUDY DESIGN

This will be a Phase 2, multicenter, randomized, active-controlled, open-label study with a 3-arm parallel design, conducted at investigator sites in the United States. A total of 565 infants  $\geq$ 42 to  $\leq$ 98 days of age at the time of consent will be enrolled and randomized in a 1:1:1 ratio to receive a vaccine series with:

- c7vPnC coadministered with Prevnar 13 (Group 1 coadministration);
- c7vPnC given 1 month after Prevnar 13 (Group 2 staggered administration); or
- Prevnar 13 alone as the active control group (Group 3 control with Supplemental Dose). A single dose of c7vPnC will be administered after the Prevnar 13 series is completed in this group.

In all groups, Prevnar 13 will be administered at 2, 4, 6, and 12 months of age. c7vPnC will be administered at 2, 4, 6, and 12 months of age in Group 1; at 3, 5, 7, and 13 months of age in Group 2; and at 13 months of age in Group 3. **Note:** In this document, and related study documents, vaccine (investigational product) Doses 1, 2, 3, and 4 specifically refer to the doses of c7vPnC administered in Groups 1 and 2, or the doses of Prevnar 13 administered in the control group (Group 3). The dose of c7vPnC administered in Group 3 will be referred to as the Supplemental Dose. See Table 1 for a summary of study groups and key procedures.

 Table 1.
 Summary of Study Groups and Key Procedures

| | 2<br>mo/o | 3<br>mo/o | 4<br>mo/o | 5<br>mo/o | 6<br>mo/o | 7<br>mo/o | 8<br>mo/o | 12<br>mo/o | 13<br>mo/o | 14<br>mo/o | 18<br>mo/o | 19<br>mo/o |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Group 1 Coadmin. | c7vPnC<br>Dose 1 | | c7vPnC<br>Dose 2 | | c7vPnC<br>Dose 3 | Blood<br>draw | | Blood<br>draw | Blood<br>draw | | Phone contact | |
| c7vPnC<br>(n= ~188) | Prev13 | | Prev13 | | Prev13 | | | c7vPnC<br>Dose 4<br>Prev13 | | | | |
| Group 2 Staggered c7vPnC (n= ~188) | Prev13 | c7vPnC<br>Dose 1 | Prev13 | c7vPnC<br>Dose 2 | Prev13 | Blood<br>draw<br>c7vPnC<br>Dose 3 | Blood<br>draw | Prev13 | Blood<br>draw<br>c7vPnC<br>Dose 4 | Blood<br>draw | | Phone contact |
| Group 3 Control (n= ~188) | Prev13<br>Dose 1 | | Prev13<br>Dose 2 | | Prev13<br>Dose 3 | Blood<br>draw | | Blood<br>draw<br>Prev13<br>Dose 4 | Blood<br>draw<br>c7vPnC<br>Suppl.<br>Dose | CCI | | Phone contact |

Abbreviations: Coadmin. = coadministered; mo/o = months old; Prev13 = Prevnar 13; Suppl. = supplemental.

Vaccine containing diphtheria, tetanus, and acellular pertussis antigens will be administered at 2, 4, and 6 months of age. This is as part of routine standard of care in the United States,

Other routine pediatric vaccines may be administered in this study, with or without certain restrictions.

Subjects will be observed for 30 minutes after each dose of c7vPnC in Groups 1 and 2, and after Prevnar 13 and the Supplemental Dose of c7vPnC in Group 3. In all groups, prompted local reactions (pain, redness, and swelling at the injection site), systemic events (fever, decreased appetite, drowsiness/increased sleep, and irritability), and use of antipyretic/pain medications occurring within 7 days after Doses 1 to 4 and the Supplemental Dose will be collected each day in the electronic diary (e-diary). SAEs and NDCMCs will be collected for the entire duration of the study. AEs (including nonserious AEs, SAEs, and NDCMCs) will be collected from the signing of the informed consent document to 1 month after Dose 3 and from Dose 4 to 1 month after Dose 4 or 1 month after the Supplemental Dose in Group 3. Approximately 6 months after Dose 4 or the Supplemental Dose, the sites will contact the subject's legally acceptable representative via telephone to inquire about SAEs and NDCMCs. Blood will be drawn for immunogenicity assessments 1 month after Dose 3, prior to receipt of Dose 4, and 1 month after Dose 4



#### 3.1. Duration of Subject Participation

Each subject will participate in the study for approximately 16 to 17 months.

#### 3.2. Duration of Study

The study duration is estimated to be approximately 25 months.

## 3.3. Number of Subjects

A total of 565 subjects will be randomized (approximately 188 subjects per arm). Assuming a 15% dropout rate at the time of Dose 3, approximately 160 subjects per arm would be evaluable for immunogenicity. Subjects who withdraw or are withdrawn from the study after randomization will not be replaced, regardless of the reason for withdrawal.

#### 4. SUBJECT ELIGIBILITY CRITERIA

This study can fulfill its objectives only if appropriate subjects are enrolled. The following eligibility criteria are designed to select subjects for whom participation in the study is considered appropriate. All relevant medical and nonmedical conditions should be taken into consideration when deciding whether a particular subject is suitable for this protocol.

Subject eligibility should be reviewed and documented by an appropriate member of the investigator's study team before subjects are included in the study.

#### 4.1. Inclusion Criteria

Subjects must meet all of the following inclusion criteria to be eligible for enrollment into the study:

- 1. Evidence of a personally signed and dated informed consent document indicating that the subject's legally acceptable representative has been informed of all pertinent aspects of the study.
- 2. Subjects whose legally acceptable representative is willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
- 3. Male or female infant born at >36 weeks of gestation and aged 2 months ( $\ge$ 42 to  $\le$ 98 days) at the time of consent (the day of birth is considered day of life 1).
- 4. Healthy infant determined by medical history, physical examination, and clinical judgment.
- 5. Expected to be available for the duration of the study and whose legally acceptable representative can be contacted by telephone during study participation.

#### 4.2. Exclusion Criteria

Subjects with any of the following characteristics/conditions will not be included in the study:

- 1. Subjects who are direct descendants (child or grandchild) of: investigational site staff members directly involved in the conduct of the study; site staff members otherwise supervised by the investigator; or Pfizer employees directly involved in the conduct of the study.
- 2. Previous vaccination with licensed or investigational pneumococcal vaccine.
- 3. Prior receipt of routine pediatric vaccines, with the exception of hepatitis B vaccine.
- 4. Previous receipt of >1 dose of hepatitis B vaccine.
- 5. Prior receipt of hepatitis B vaccine at age  $\geq$ 30 days.

- 6. Contraindication to immunization with diphtheria, tetanus, pertussis, or 13-valent pneumococcal conjugate vaccines, according to each vaccine's product information.
- 7. History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of the investigational product or any diphtheria toxoid-containing vaccine.
- 8. History of microbiologically proven invasive disease caused by *S pneumoniae*.
- 9. Major known congenital malformation or serious chronic disorder.
- 10. Significant neurological disorder or history of seizure including febrile seizure, or significant stable or evolving disorders such as cerebral palsy, encephalopathy, hydrocephalus, or other significant disorders. Does not include resolving syndromes due to birth trauma, such as Erb's palsy and/or hypotonic-hyporesponsive episodes.
- 11. Other acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
- 12. Subjects who receive treatment with immunosuppressive therapy, including cytotoxic agents or systemic corticosteroids, or planned receipt through the last study visit. If systemic corticosteroids have been administered short term (<14 days) for treatment of an acute illness, subjects should not be enrolled into the study until corticosteroid therapy has been discontinued for at least 28 days before investigational product administration. Inhaled/nebulized, intra-articular, intrabursal, or topical (skin, eyes, or ears) corticosteroids are permitted.
- 13. Subjects with known or suspected immunodeficiency or other conditions associated with immunosuppression, including, but not limited to, immunoglobulin class/subclass deficiencies, DiGeorge syndrome, generalized malignancy, human immunodeficiency virus infection, leukemia, lymphoma, or organ or bone marrow transplant.
- 14. Bleeding diathesis or condition associated with prolonged bleeding time that would in the opinion of the investigator contraindicate intramuscular injection.
- 15. Receipt of blood/plasma products or immunoglobulins (including hepatitis B immunoglobulin) since birth, or planned receipt through the last study visit.
- 16. Participation in other studies involving investigational drug(s) or interventional studies or receipt of any other investigational vaccines, drugs, or medical devices prior to study entry and/or during study participation. Participation in purely observational studies is acceptable.

#### 4.3. Temporary Delay Criteria

The following conditions are temporary or self-limiting and a subject may be vaccinated and/or have blood drawn at the visit once the condition(s) has/have resolved and no other exclusion criteria are met. The blood draw prior to Dose 3 (in Group 2 only) and prior to Dose 4/Supplemental Dose should take place on the same day as the administration of investigational product.

# 4.3.1. Criteria for Temporarily Delaying Dose Administration (Doses 1, 2, 3, and 4 and the Supplemental Dose)

- Febrile illness (eg, rectal temperature ≥100.4°F [≥38°C]) or other acute illness within 48 hours before each dose.
- Receipt of any inactivated vaccine within 14 days or any live vaccine within 28 days before each dose.
- Receipt of short-term (<14 days) systemic corticosteroids. Dose administration should be delayed until systemic corticosteroid use has been discontinued for at least 28 days (inhaled/nebulized, intra-articular, intrabursal, or topical [skin, eyes, or ears] corticosteroids are permitted).

# 4.3.2. Criteria for Temporarily Delaying Blood Draw (Prior to Dose 3, 1 Month After Dose 3, Prior to Dose 4, and 1 Month After Dose 4 and the Supplemental Dose)

• Receipt of antibiotic therapy within 72 hours before blood draw.

#### 4.4. Sponsor's Qualified Medical Personnel

The contact information for the sponsor's appropriately qualified medical personnel for the study is documented in the study contact list located in the supporting study documentation.

To facilitate access to appropriately qualified medical personnel on study-related medical questions or problems, the subject's legally acceptable representative is provided with a contact card. The contact card contains, at a minimum, protocol and investigational product identifiers, subject study numbers, contact information for the investigator site, and contact details for a contact center in the event that the investigator site staff cannot be reached to provide advice on a medical question or problem originating from another healthcare professional not involved in the subject's participation in the study. The contact number can also be used by investigator staff if they are seeking advice on medical questions or problems; however, it should be used only in the event that the established communication pathways between the investigator site and the study team are not available. It is therefore intended to augment, but not replace, the established communication pathways between the investigator site and the study team for advice on medical questions or problems that may arise during the study. The contact number is not intended for use by the subject's legally acceptable representative directly, and if the subject's legally acceptable representative calls that number, he or she will be directed back to the investigator site.

#### 5. INVESTIGATIONAL PRODUCTS

For the purposes of this study, and per International Council for Harmonisation (ICH) guidelines, investigational product is defined as a pharmaceutical form of an active ingredient or placebo being tested or used as a reference/comparator in a clinical trial, including a product with a marketing authorization when used or assembled (formulated or packaged) in a way different from the approved form, or when used for an unapproved indication, or when used to gain further information about an approved use (ICH E6 1.33).

For this study, the investigational products are c7vPnC and Prevnar 13.

## 5.1. Allocation to Investigational Product

The investigator's knowledge of the treatment should not influence the decision to enroll a particular subject or affect the order in which subjects are enrolled.

Allocation of subjects to vaccine groups will proceed through the use of an interactive response technology (IRT) system (interactive Web-based response [IWR]). The site personnel (study coordinator or specified designee) will be required to enter or select information including but not limited to the user's identification (ID) and password, the protocol number, and the subject number. The site personnel will then be provided with a randomization number and container number when investigational product is being supplied via the IRT system. The IRT system will provide a confirmation report containing the subject number, randomization number, and container number assigned. The confirmation report must be stored in the site's files.

The study-specific IRT reference manual will provide the contact information and further details on the use of the IRT system.

#### **5.2. Subject Compliance**

All doses of vaccine will be administered by the appropriately designated study staff at the investigator site.

# 5.3. Investigational Product Supplies

Study vaccines will be packed and labeled as investigational product in accordance with current guidelines and applicable local and legal regulatory requirements. The formulations of c7vPnC and Prevnar 13 are described below.

#### 5.3.1. Dosage Form(s) and Packaging

c7vPnC contains saccharides of the capsular antigens to *S pneumoniae* serotypes 8, 10A, 11A, 12F, 15B, 22F, and 33F individually conjugated to nontoxic diphtheria toxin CRM<sub>197</sub>.



Prevnar 13 contains saccharides from pneumococcal serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F individually conjugated to nontoxic diphtheria toxin CRM<sub>197</sub>. The vaccine is a sterile suspension formulated to contain 2.2  $\mu$ g of each saccharide, except for 4.4  $\mu$ g of 6B, per 0.5-mL dose. The vaccine contains 295  $\mu$ g succinate buffer, 0.85% sodium chloride, 100  $\mu$ g polysorbate 80, 0.125 mg aluminum as aluminum phosphate, and 34  $\mu$ g CRM<sub>197</sub>, per 0.5-mL dose.<sup>68</sup>

c7vPnC and Prevnar 13 will be supplied to the site as packaged single-use prefilled syringes and labeled according to local regulatory requirements.

#### 5.3.2. Preparation and Dispensing

See the Investigational Product Manual (IP manual) for instructions on how to prepare c7vPnC and Prevnar 13 for administration. c7vPnC and Prevnar 13 should be prepared and dispensed by an appropriately qualified and experienced member of the study staff (eg, physician, nurse, physician's assistant, nurse practitioner, pharmacy assistant/technician, or pharmacist) as allowed by local, state, and institutional guidance.

#### 5.4. Administration

Investigational product, ie, c7vPnC for Groups 1 and 2 and the Supplemental Dose (Group 3), and Prevnar 13 (control) in Group 3, will be administered into the thigh of the left leg as specified below.

- Group 1: Each dose (0.5 mL) of c7vPnC will be administered intramuscularly (IM) into the anterolateral thigh muscle of the left leg and each dose (0.5 mL) of Prevnar 13 will be administered IM into the anterolateral thigh muscle of the right leg.
- Group 2: Each dose (0.5 mL) of Prevnar 13 (given 1 month before the c7vPnC dose) will be administered IM into the anterolateral thigh muscle of the right leg and each dose (0.5 mL) of c7vPnC will be administered IM into the anterolateral thigh muscle of the left leg.
- Group 3: Prevnar 13 (0.5 mL) and the Supplemental Dose of c7vPnC will be administered IM into the anterolateral thigh muscle of the left leg.

Other permitted routine pediatric injectable vaccines (including diphtheria, tetanus, and acellular pertussis [DTaP]-containing vaccines) must be administered in a different limb from the site of administration of c7vPnC in Groups 1 and 2 or Prevnar 13/c7vPnC Supplemental Dose in Group 3. Concomitant injectable vaccines will be administered with Prevnar 13 (not c7vPnC) in Group 2. The location of the injection of each vaccine administered (investigational product and other) will be recorded.

Standard vaccination practices must be observed and vaccine must not be injected into blood vessels. Appropriate medication and other supportive measures for management of an acute hypersensitivity reaction should be available in accordance with local guidelines for standard immunization practices.

Administration of vaccines in this study should be performed by an appropriately qualified, Good Clinical Practice (GCP)-trained, and vaccine-experienced member of the study staff (eg, physician, nurse, physician's assistant, nurse practitioner, pharmacist, or medical assistant) as allowed by local, state, and institutional guidance.

Vaccine administration details will be recorded on the case report form (CRF).

#### 5.5. Investigational Product Storage

The investigator or an approved representative, eg, pharmacist, will ensure that all investigational products, including any comparator and/or marketed products, are stored in a secured area with controlled access under required storage conditions and in accordance with applicable regulatory requirements.

Investigational products should be stored in their original containers and in accordance with the labels.

Investigational products will be shipped to the study site after required regulatory and legal documents have been received by the sponsor.



Any storage conditions stated in the SRSD will be superseded by the storage conditions stated on the product label.

Site systems must be capable of measuring and documenting (for example, via a log), at a minimum, daily minimum and maximum temperatures for all site storage locations (as applicable, including frozen, refrigerated, and/or room-temperature products). This should be captured from the time of investigational product receipt throughout the study. Even for continuous-monitoring systems, a log or site procedure that ensures active evaluation for excursions should be available. The intent is to ensure that the minimum and maximum temperature is checked each business day to confirm that no excursion occurred since the last evaluation and to provide the site with the capability to store or view the minimum/maximum temperature for all nonworking days upon return to normal operations. The operation of the temperature-monitoring device and storage unit (for example, refrigerator), as applicable, should be regularly inspected to ensure they are maintained in working order.

Any excursions from the product label storage conditions should be reported to Pfizer upon discovery. The site should actively pursue options for returning the product to the storage conditions described in the labeling, as soon as possible. Deviations from the storage requirements, including any actions taken, must be documented and reported to Pfizer.

Once an excursion is identified, the investigational product must be quarantined and not used until Pfizer provides permission to use the investigational product. It will not be considered a protocol deviation if Pfizer approves the use of the investigational product after the

temperature excursion. Use of the investigational product prior to Pfizer approval will be considered a protocol deviation. Specific details regarding information the site should report for each excursion will be provided to the site.

Receipt of materials, door opening and closing, and other routine handling operations where the products are briefly out of the temperature range described in the labeling are not considered excursions.

#### 5.6. Investigational Product Accountability

The investigator site must maintain adequate records documenting the receipt, use, loss, or other disposition of the investigational product supplies. All investigational products will be accounted for using a drug accountability form/record.

Used needles and syringes should be disposed of according to local practice. Empty outer investigational product containers must be retained until reviewed by the sponsor's site staff and then may be destroyed after the sponsor's site staff has performed accountability. Investigational product return/destruction must be documented on the accountability log.

#### 5.6.1. Destruction of Investigational Product Supplies

The sponsor or designee will provide guidance on the destruction of unused investigational product (eg, at the site). If destruction is authorized to take place at the investigator site, the investigator must ensure that the materials are destroyed in compliance with applicable environmental regulations, institutional policy, and any special instructions provided by Pfizer, and all destruction must be adequately documented.

#### 5.7. Concomitant Vaccines/Medications

#### 5.7.1. Concomitant Vaccines to Be Administered at Study Visits

DTaP-containing vaccine (in combination with other antigens, such as polio) will be administered concomitantly at 2, 4, and 6 months of age.

All vaccines administered will be recorded in the CRFs.

#### 5.7.2. Prohibited Vaccines/Medications During the Study

- Receipt of any investigational vaccines, drugs, or medical devices is prohibited during subject participation in the study.
- Receipt of any nonstudy pneumococcal vaccine is prohibited during subject participation in the study.
- Receipt of blood/plasma products, immunoglobulins, and/or immunosuppressive therapy (including a ≥14-day course of systemic corticosteroids) is prohibited during subject participation in the study.

#### 5.7.3. Permitted Vaccines/Medications During the Study

- If not in the DTaP-combination vaccine, polio, hepatitis B, and *Haemophilus influenzae* type b vaccines may be given at 2, 4, and 6 months of age.
- Measles, mumps, and rubella (MMR) vaccine may be administered concomitantly at 12 months of age or according to the permitted treatment windows for other nonprohibited licensed vaccines below.
- Rotavirus vaccine may be given at any time throughout the study.
- Receipt of quadrivalent meningococcal conjugate vaccine is permitted during the study only after blood is collected at the visit occurring 1 month after Dose 4
- Other nonprohibited licensed vaccines may be given between the blood draw 1 month after Dose 3 and 14 days before Dose 4 for inactivated vaccines or 28 days before Dose 4 for live vaccines, according to local or national recommendations. Following the blood draw performed 1 month after Dose 4 CCI all licensed vaccines are permitted.
- Licensed inactivated influenza vaccine may be given to eligible study subjects during influenza season.
- Use of a topical anesthetic is permitted.
- The use of prophylactic antipyretic/pain medication, while permitted, is not recommended on the day of investigational product administration (before or after vaccination).
- Inhaled/nebulized, topical (skin, eyes or ears), or localized injections of corticosteroids (eg, intra-articular or intrabursal administration) are permitted during subject participation in the study.
- Prescription and nonprescription medications, vitamins, minerals, and herbal remedies are permitted during subject participation in the study.

#### 5.7.4. Recording Prior and Concomitant Treatments

The name and date of administration for all vaccinations should be collected from the time of signing of the informed consent document to 1 month after Dose 4/Supplemental Dose and will be recorded in the CRF. At Visit 1, information on prior vaccinations will also be recorded in the CRF.

Concomitant medications used to treat an NDCMC or SAE should be collected from the signing of informed consent through 6 months after Dose 4/Supplemental Dose (telephone contact) and will be recorded in the CRF.

#### 6. STUDY PROCEDURES

The study procedures described by assigned group are provided below and summarized in the Schedule of Activities. The day of the first investigational product vaccination is considered to be Day 1.

Prior to randomization, all subjects undergo the same procedures.

#### 6.1. Group 1 (Coadministration) Study Procedures

#### 6.1.1. Group 1 Visit 1 (Dose 1: 2-Month Visit, Day 1)

Prior to randomization:

- A personally signed and dated informed consent document indicating that the subject's legally acceptable representative has been informed of all pertinent aspects of the study before performing any study-specific procedures.
- Record the subject's demographic information (including date of birth, sex, race, and ethnicity).
- Obtain and record the subject's medical history including prior vaccinations.
- Perform physical examination evaluating any clinically significant abnormalities within the following body systems: general appearance; skin; head, eyes, ears, nose, and throat; heart; lungs; abdomen; musculoskeletal; extremities; neurological; and lymph nodes. Clinically significant abnormal results will be recorded in the CRF.
- Measure and record the subject's rectal temperature (°F/°C).
- Ensure that all inclusion criteria, none of the exclusion criteria, and none of the temporary delay criteria are met.
- Assign randomization number and investigational product container numbers via the IRT. This must be the last step before proceeding. A site staff member will prepare the investigational product according to the IP manual.

#### After randomization:

- Administer a single 0.5-mL injection of c7vPnC into the left anterolateral thigh and a single 0.5-mL injection of Prevnar 13 into the right anterolateral thigh.
- Administer DTaP-containing vaccine and other permitted vaccines (to be administered into a limb other than the site of c7vPnC injection).
- Site staff will observe the subject for at least 30 minutes after vaccination for any acute reactions. Record any AEs on the CRF and on an SAE form as applicable. Record concomitant medications used to treat SAEs and NDCMCs.

- Issue the subject's legally acceptable representative a measuring device to measure injection site reactions and a digital thermometer and provide instructions on their use.
- Issue the subject's legally acceptable representative an e-diary (device or application). Provide instructions on use and completion of the e-diary. Ask the subject's legally acceptable representative to complete the e-diary from Day 1 to Day 7, with Day 1 being the day of vaccination.
- Ask the subject's legally acceptable representative to contact the investigator site staff or investigator as soon as possible during the 7-day postvaccination period if the subject has a fever >104.0°F (>40.0°C), redness and/or swelling at the injection site measuring >14 measuring device units (>7 cm), or severe injection site pain (causes limitation of limb movement) to determine if the event requires further assessment by the investigator.
- Ask the subject's legally acceptable representative to contact the investigator or investigator site staff as soon as possible if any significant illness or medical event (eg, emergency room visit or hospitalization) occurs.
- Inform the subject's legally acceptable representative that use of prophylactic antipyretic/pain medication, while permitted, is not recommended on the day of investigational product administration (before or after vaccination).
- The investigator or an authorized designee completes the CRF and updates the investigational product accountability records.

#### 6.1.2. Group 1 Visit 2 (Dose 2: 4-Month Visit, 42 to 63 Days After Dose 1)

- Ensure and document that the subject continues to be eligible for the study (see Section 6.5 for withdrawal information), and none of the temporary delay criteria are met.
- Record vaccines administered since Visit 1 as described in Section 5.7.4.
- Review the subject's e-diary data with the subject's legally acceptable representative; collect stop dates of any e-diary events ongoing on the last day that the e-diary was completed and record stop dates in the CRF.
- Determine whether any AEs (includes nonserious AEs, SAEs, and NDCMCs) have
  occurred since the previous visit and follow up on any previously reported events to
  determine the outcome (ie, record stop dates or confirm if they are still continuing) and
  record as described in Section 8, and record concomitant medications used to treat SAEs
  and NDCMCs.
- Measure and record the subject's rectal temperature ( ${}^{\circ}F/{}^{\circ}C$ ).
- Administer a single 0.5-mL injection of c7vPnC into the left anterolateral thigh and a single 0.5-mL injection of Prevnar 13 into the right anterolateral thigh.
• Administer DTaP-containing vaccine and other permitted vaccines (to be administered into a limb other than the site of c7vPnC injection).

#### After vaccination:

- Site staff will observe the subject for at least 30 minutes after vaccination for any acute reactions. Record any AEs on the CRF and on an SAE form as applicable. Record concomitant medications used to treat SAEs and NDCMCs.
- Confirm that the e-diary is working and review instructions if necessary. Remind the subject's legally acceptable representative to complete the e-diary from Day 1 to Day 7, with Day 1 being the day of vaccination. Provide thermometer or measuring device if needed.
- Ask the subject's legally acceptable representative to contact the investigator site staff or investigator as soon as possible during the 7-day postvaccination period if the subject experiences fever >104.0°F (>40.0°C), redness or swelling at the injection site measuring >14 measuring device units (>7 cm), or severe injection site pain (causes limitation of limb movement) to determine if the event requires further assessment by the investigator.
- Remind the subject's legally acceptable representative to contact the investigator or investigator site staff as soon as possible if any significant illness or medical event (eg, emergency room visit or hospitalization) occurs during the study period.
- Remind the subject's legally acceptable representative that use of prophylactic antipyretic/pain medication, while permitted, is not recommended on the day of investigational product administration (before or after vaccination).
- The investigator or an authorized designee completes the CRF and updates the investigational product accountability records.

## 6.1.3. Group 1 Visit 3 (Dose 3: 6-Month Visit, 42 to 63 Days After Dose 2)

- Ensure and document that the subject continues to be eligible for the study (see Section 6.5 for withdrawal information), and none of the temporary delay criteria are met.
- Record vaccines administered since Visit 2 as described in Section 5.7.4.
- Review the subject's e-diary data with the subject's legally acceptable representative; collect stop dates of any e-diary events ongoing on the last day that the e-diary was completed and record stop dates in the CRF.
- Determine whether any AEs (includes nonserious AEs, SAEs, and NDCMCs) have occurred since the previous visit and follow up on any previously reported events to determine the outcome (ie, record stop dates or confirm if they are still continuing) and record as described in Section 8, and record concomitant medications used to treat SAEs and NDCMCs.

- Measure and record the subject's rectal temperature (°F/°C).
- Administer a single 0.5-mL injection of c7vPnC into the left anterolateral thigh and a single 0.5-mL injection of Prevnar 13 into the right anterolateral thigh.
- Administer DTaP-containing vaccine and other permitted vaccines (to be administered into a limb other than the site of c7vPnC injection).

### After vaccination:

- Site staff will observe the subject for at least 30 minutes after vaccination for any acute reactions. Record any AEs on the CRF and on an SAE form as applicable. Record concomitant medications used to treat SAEs and NDCMCs.
- Confirm that the e-diary is working and review instructions if necessary. Remind the subject's legally acceptable representative to complete the e-diary from Day 1 to Day 7, with Day 1 being the day of vaccination. Provide thermometer or measuring device if needed.
- Ask the subject's legally acceptable representative to contact the investigator site staff or investigator as soon as possible during the 7-day postvaccination period if the subject experiences fever >104.0°F (>40.0°C), redness or swelling at the injection site measuring >14 measuring device units (>7 cm), or severe injection site pain (causes limitation of limb movement) to determine if the event requires further assessment by the investigator.
- Remind the subject's legally acceptable representative to contact the investigator or investigator site staff as soon as possible if any significant illness or medical event (eg, emergency room visit or hospitalization) occurs during the study period.
- Remind the subject's legally acceptable representative that use of prophylactic antipyretic/pain medication, while permitted, is not recommended on the day of investigational product administration (before or after vaccination).
- The investigator or an authorized designee completes the CRF and updates the investigational product accountability records.

## 6.1.4. Group 1 Visit 4 (Follow-up: 7-Month Visit, 28 to 42 Days After Dose 3)

- Ensure and document that the subject continues to be eligible for the study (see Section 6.5 for withdrawal information), and none of the temporary delay criteria are met.
- Record vaccines administered since Visit 3 as described in Section 5.7.4.
- Review the subject's e-diary data with the subject's legally acceptable representative; collect stop dates of any e-diary events ongoing on the last day that the e-diary was completed and record stop dates in the CRF.

- Collect the e-diary (if device provided).
- Determine whether any AEs (includes nonserious AEs, SAEs, and NDCMCs) have
  occurred since the previous visit and follow up on any previously reported events to
  determine the outcome (ie, record stop dates or confirm if they are still continuing) and
  record as described in Section 8, and record concomitant medications used to treat SAEs
  and NDCMCs.
- Collect a blood sample of approximately 5 mL for immunogenicity (a topical anesthetic is permitted).
- Remind the subject's legally acceptable representative to contact the investigator or investigator site staff as soon as possible if any significant illness or medical event (eg, emergency room visit or hospitalization) occurs during the study period.
- Remind the subject's legally acceptable representative that use of prophylactic antipyretic/pain medication, while permitted, is not recommended on the day of investigational product administration (before or after vaccination).
- The investigator or an authorized designee completes the CRF.

## 6.1.5. Group 1 Visit 5 (Dose 4: 12-Month Visit, 365 to 386 Days of Age)

- Ensure and document that the subject continues to be eligible for the study (see Section 6.5 for withdrawal information), and none of the temporary delay criteria are met.
- Record vaccines administered since Visit 4 as described in Section 5.7.4.
- Determine whether any SAEs or NDCMCs have occurred since the previous visit and follow up on any previously reported events to determine the outcome (ie, record stop dates or confirm if they are still continuing) and record as described in Section 8, and record concomitant medications used to treat SAEs and NDCMCs.
- Measure and record the subject's rectal temperature ( ${}^{\circ}F/{}^{\circ}C$ ).
- Collect a blood sample of approximately 5 mL for immunogenicity prior to vaccination (a topical anesthetic is permitted).
- Administer a single 0.5-mL injection of c7vPnC into the left anterolateral thigh and a single 0.5-mL injection of Prevnar 13 into the right anterolateral thigh.
- Administer permitted vaccines (to be administered into a limb other than the site of c7vPnC injection).

#### After vaccination:

- Site staff will observe the subject for at least 30 minutes after vaccination for any acute reactions. Record any AEs on the CRF and on an SAE form as applicable. Record concomitant medications used to treat SAEs and NDCMCs.
- Issue the subject's legally acceptable representative an e-diary (if device needed). Provide and review instructions on use and completion of the e-diary. Ask the subject's legally acceptable representative to complete the e-diary from Day 1 to Day 7, with Day 1 being the day of vaccination. Provide thermometer or measuring device if needed.
- Ask the subject's legally acceptable representative to contact the investigator site staff or investigator immediately during the 7-day postvaccination period if the subject experiences fever >104.0°F (>40.0°C), redness or swelling at the injection site measuring >14 measuring device units (>7 cm), or severe injection site pain (causes limitation of limb movement) to determine if the event requires further assessment by the investigator.
- Remind the subject's legally acceptable representative to contact the investigator or investigator site staff as soon as possible if any significant illness or medical event (eg, emergency room visit or hospitalization) occurs.
- Remind the subject's legally acceptable representative that use of prophylactic antipyretic/pain medication, while permitted, is not recommended on the day of investigational product administration (before or after vaccination).
- The investigator or an authorized designee completes the CRF and updates the investigational product accountability records.

## 6.1.6. Group 1 Visit 6 (Follow-up: 13-Month Visit, 28 to 42 Days After Dose 4)

- Ensure and document that the subject continues to be eligible for the study (see Section 6.5 for withdrawal information), and none of the temporary delay criteria are met.
- Record vaccines administered since Visit 5 as described in Section 5.7.4.
- Review the subject's e-diary data with the subject's legally acceptable representative; collect stop dates of any e-diary events ongoing on the last day that the e-diary was completed and record stop dates in the CRF.
- Collect the e-diary (if device provided).
- Determine whether any AEs (includes nonserious AEs, SAEs, or NDCMCs) have occurred since the previous visit and follow up on any previously reported events to determine the outcome (ie, record stop dates or confirm if they are still continuing) and record as described in Section 8, and record concomitant medications used to treat SAEs and NDCMCs.

- Collect a blood sample of approximately 5 mL for immunogenicity assessments (a topical anesthetic is permitted).
- Remind the subject's legally acceptable representative to contact the investigator or investigator site staff immediately if any significant illness or medical event (eg, emergency room visit or hospitalization) occurs.
- The investigator or an authorized designee completes the CRF.

# 6.1.7. Group 1 Visit 7 (Follow-up: 18-Month Phone Contact, 168 to 196 Days After Dose 4)

- Contact the subject's legally acceptable representative by telephone approximately 6 months after the last dose of c7vPnC; this contact should be attempted for all subjects who have received at least 1 dose of c7vPnC, unless the subject's legally acceptable representative has withdrawn consent.
- Determine whether any SAEs or NDCMCs have occurred since the previous visit and follow up on any previously reported events to determine the outcome (ie, record stop dates or confirm if they are still continuing) and record as described in Section 8, and record concomitant medications used to treat SAEs and NDCMCs.
- The investigator or an authorized designee completes the CRF.

## 6.2. Group 2 (Staggered Administration) Study Procedures

# 6.2.1. Group 2 Visit 1 (Prevnar 13: 2-Month Visit, Day 1)

Prior to randomization:

- A personally signed and dated informed consent document indicating that the subject's legally acceptable representative has been informed of all pertinent aspects of the study before performing any study-specific procedures.
- Record the subject's demographic information (including date of birth, sex, race, and ethnicity).
- Obtain and record the subject's medical history including prior vaccinations.
- Perform physical examination evaluating any clinically significant abnormalities within the following body systems: general appearance; skin; head, eyes, ears, nose, and throat; heart; lungs; abdomen; musculoskeletal; extremities; neurological; and lymph nodes. Clinically significant abnormal results will be recorded in the CRF.
- Ensure that all inclusion criteria and none of the exclusion criteria are met.

• Assign randomization number and investigational product container number via the IRT. This must be the last step before proceeding. A site staff member will prepare the investigational product according to the IP manual.

#### After randomization:

- Administer a single 0.5-mL injection of Prevnar 13 into the right anterolateral thigh.
- Administer DTaP-containing vaccine and other permitted vaccines (to be administered into a limb other than the left leg).
- Ask the subject's legally acceptable representative to contact the investigator or investigator site staff as soon as possible if any significant illness or medical event (eg, emergency room visit or hospitalization) occurs.
- Inform the subject's legally acceptable representative that use of prophylactic antipyretic/pain medication, while permitted, is not recommended on the day of investigational product administration (before or after vaccination).
- The investigator or an authorized designee completes the CRF and updates the investigational product accountability records.

# 6.2.2. Group 2 Visit 2 (c7vPnC Dose 1: 3-Month Visit, 21 to 35 Days After Prevnar 13 at Visit 1)

- Ensure and document that the subject continues to be eligible for the study (see Section 6.5 for withdrawal information), and none of the temporary delay criteria are met.
- Record vaccines administered since Visit 1 as described in Section 5.7.4.
- Determine whether any AEs (includes nonserious AEs, SAEs, and NDCMCs) have occurred since the previous visit and follow up on any previously reported events to determine the outcome (ie, record stop dates or confirm if they are still continuing) and record as described in Section 8, and record concomitant medications used to treat SAEs and NDCMCs.
- Measure and record the subject's rectal temperature ( ${}^{\circ}F/{}^{\circ}C$ ).
- Administer a single 0.5-mL injection of c7vPnC into the left anterolateral thigh.

## After vaccination:

• Site staff will observe the subject for at least 30 minutes after vaccination for any acute reactions. Record any AEs on the CRF and on an SAE form as applicable. Record concomitant medications used to treat SAEs and NDCMCs.

- Issue the subject's legally acceptable representative a measuring device to measure injection site reactions and a digital thermometer and provide instructions on their use.
- Issue the subject's legally acceptable representative an e-diary (device or application). Provide instructions on use and completion of the e-diary. Ask the subject's legally acceptable representative to complete the e-diary from Day 1 to Day 7, with Day 1 being the day of vaccination.
- Ask the subject's legally acceptable representative to contact the investigator site staff or investigator as soon as possible during the 7-day postvaccination period if the subject has a fever >104.0°F (>40.0°C), redness and/or swelling at the injection site measuring >14 measuring device units (>7 cm), or severe injection site pain (causes limitation of limb movement) to determine if the event requires further assessment by the investigator.
- Ask the subject's legally acceptable representative to contact the investigator or investigator site staff as soon as possible if any significant illness or medical event (eg, emergency room visit or hospitalization) occurs during the study period.
- Remind the subject's legally acceptable representative that use of prophylactic antipyretic/pain medication, while permitted, is not recommended on the day of investigational product administration (before or after vaccination).
- The investigator or an authorized designee completes the CRF and updates the investigational product accountability records.

# 6.2.3. Group 2 Visit 3 (Prevnar 13: 4-Month Visit, 42 to 63 Days After Prevnar 13 at Visit 1)

- Ensure and document that the subject continues to be eligible for the study (see Section 6.5 for withdrawal information).
- Record vaccines administered since Visit 2 as described in Section 5.7.4.
- Review the subject's e-diary data with the subject's legally acceptable representative; collect stop dates of any e-diary events ongoing on the last day that the e-diary was completed and record stop dates in the CRF.
- Determine whether any AEs (includes nonserious AEs, SAEs, and NDCMCs) have occurred since the previous visit and follow up on any previously reported events to determine the outcome (ie, record stop dates or confirm if they are still continuing) and record as described in Section 8, and record concomitant medications used to treat SAEs and NDCMCs.
- Administer a single 0.5-mL injection of Prevnar 13 into the right anterolateral thigh.
- Administer DTaP-containing vaccine and other permitted vaccines (to be administered into a limb other than the left leg).

#### After vaccination:

- Remind the subject's legally acceptable representative to contact the investigator or investigator site staff as soon as possible if any significant illness or medical event (eg, emergency room visit or hospitalization) occurs during the study period.
- Remind the subject's legally acceptable representative that use of prophylactic antipyretic/pain medication, while permitted, is not recommended on the day of investigational product administration (before or after vaccination).
- The investigator or an authorized designee completes the CRF and updates the investigational product accountability records.

# 6.2.4. Group 2 Visit 4 (c7vPnC Dose 2: 5-Month Visit, 21 to 35 Days After Prevnar 13 at Visit 3)

- Ensure and document that the subject continues to be eligible for the study (see Section 6.5 for withdrawal information), and none of the temporary delay criteria are met.
- Record vaccines administered since Visit 3 as described in Section 5.7.4.
- Determine whether any AEs (includes nonserious AEs, SAEs, and NDCMCs) have occurred since the previous visit and follow up on any previously reported events to determine the outcome (ie, record stop dates or confirm if they are still continuing) and record as described in Section 8, and record concomitant medications used to treat SAEs and NDCMCs.
- Measure and record the subject's rectal temperature ( ${^{\circ}F/^{\circ}C}$ ).
- Administer a single 0.5-mL injection of c7vPnC into the left anterolateral thigh.

- Site staff will observe the subject for at least 30 minutes after vaccination for any acute reactions. Record any AEs on the CRF and on an SAE form as applicable. Record concomitant medications used to treat SAEs and NDCMCs.
- Confirm that the e-diary is working and review instructions if necessary. Remind the subject's legally acceptable representative to complete the e-diary from Day 1 to Day 7, with Day 1 being the day of vaccination. Provide thermometer or measuring device if needed.
- Ask the subject's legally acceptable representative to contact the investigator site staff or investigator as soon as possible during the 7-day postvaccination period if the subject experiences fever >104.0°F (>40.0°C), redness or swelling at the injection site measuring >14 measuring device units (>7 cm), or severe injection site pain (causes limitation of limb movement) to determine if the event requires further assessment by the investigator.

- Remind the subject's legally acceptable representative to contact the investigator or investigator site staff as soon as possible if any significant illness or medical event (eg, emergency room visit or hospitalization) occurs during the study period.
- Remind the subject's legally acceptable representative that use of prophylactic antipyretic/pain medication, while permitted, is not recommended on the day of investigational product administration (before or after vaccination).
- The investigator or an authorized designee completes the CRF and updates the investigational product accountability records.

# 6.2.5. Group 2 Visit 5 (Prevnar 13: 6-Month Visit, 42 to 63 Days After Prevnar 13 at Visit 3)

- Ensure and document that the subject continues to be eligible for the study (see Section 6.5 for withdrawal information).
- Record vaccines administered since Visit 4 as described in Section 5.7.4.
- Review the subject's e-diary data with the subject's legally acceptable representative; collect stop dates of any e-diary events ongoing on the last day that the e-diary was completed and record stop dates in the CRF.
- Determine whether any AEs (includes nonserious AEs, SAEs, and NDCMCs) have occurred since the previous visit and follow up on any previously reported events to determine the outcome (ie, record stop dates or confirm if they are still continuing) and record as described in Section 8, and record concomitant medications used to treat SAEs and NDCMCs.
- Administer a single 0.5-mL injection of Prevnar 13 into the right anterolateral thigh.
- Administer DTaP-containing vaccine and other permitted vaccines (to be administered into a limb other than the left leg).

- Remind the subject's legally acceptable representative to contact the investigator or investigator site staff as soon as possible if any significant illness or medical event (eg, emergency room visit or hospitalization) occurs during the study period.
- Remind the subject's legally acceptable representative that use of prophylactic antipyretic/pain medication, while permitted, is not recommended on the day of investigational product administration (before or after vaccination).
- The investigator or an authorized designee completes the CRF and updates the investigational product accountability records.

# 6.2.6. Group 2 Visit 6 (c7vPnC Dose 3: 7-Month Visit, 21 to 35 Days After Prevnar 13 at Visit 5)

- Ensure and document that the subject continues to be eligible for the study (see Section 6.5 for withdrawal information), and none of the temporary delay criteria are met.
- Record vaccines administered since Visit 5 as described in Section 5.7.4.
- Determine whether any AEs (includes nonserious AEs, SAEs, and NDCMCs) have occurred since the previous visit and follow up on any previously reported events to determine the outcome (ie, record stop dates or confirm if they are still continuing) and record as described in Section 8, and record concomitant medications used to treat SAEs and NDCMCs.
- Measure and record the subject's rectal temperature ( ${}^{\circ}F/{}^{\circ}C$ ).
- Collect a blood sample of approximately 5 mL for immunogenicity prior to vaccination (a topical anesthetic is permitted).
- Administer a single 0.5-mL injection of c7vPnC into the left anterolateral thigh.

- Site staff will observe the subject for at least 30 minutes after vaccination for any acute reactions. Record any AEs on the CRF and on an SAE form as applicable. Record concomitant medications used to treat SAEs and NDCMCs.
- Confirm that the e-diary is working and review instructions if necessary. Remind the subject's legally acceptable representative to complete the e-diary from Day 1 to Day 7, with Day 1 being the day of vaccination. Provide thermometer or measuring device if needed.
- Ask the subject's legally acceptable representative to contact the investigator site staff or investigator as soon as possible during the 7-day postvaccination period if the subject experiences fever >104.0°F (>40.0°C), redness or swelling at the injection site measuring >14 measuring device units (>7 cm), or severe injection site pain (causes limitation of limb movement) to determine if the event requires further assessment by the investigator.
- Remind the subject's legally acceptable representative to contact the investigator or investigator site staff as soon as possible if any significant illness or medical event (eg, emergency room visit or hospitalization) occurs during the study period.
- Remind the subject's legally acceptable representative that use of prophylactic antipyretic/pain medication, while permitted, is not recommended on the day of investigational product administration (before or after vaccination).

• The investigator or an authorized designee completes the CRF and updates the investigational product accountability records.

# 6.2.7. Group 2 Visit 7 (Follow-up: 8-Month Visit, 28 to 42 Days After Dose 3)

- Ensure and document that the subject continues to be eligible for the study (see Section 6.5 for withdrawal information), and none of the temporary delay criteria are met.
- Record vaccines administered since Visit 6 as described in Section 5.7.4.
- Review the subject's e-diary data with the subject's legally acceptable representative; collect stop dates of any e-diary events ongoing on the last day that the e-diary was completed and record stop dates in the CRF.
- Collect the e-diary (if device provided).
- Determine whether any AEs (includes nonserious AEs, SAEs, and NDCMCs) have
  occurred since the previous visit and follow up on any previously reported events to
  determine the outcome (ie, record stop dates or confirm if they are still continuing) and
  record as described in Section 8, and record concomitant medications used to treat SAEs
  and NDCMCs.
- Collect a blood sample of approximately 5 mL for immunogenicity (a topical anesthetic is permitted).
- Remind the subject's legally acceptable representative to contact the investigator or investigator site staff as soon as possible if any significant illness or medical event (eg, emergency room visit or hospitalization) occurs during the study period.
- Remind the subject's legally acceptable representative that use of prophylactic antipyretic/pain medication, while permitted, is not recommended on the day of investigational product administration (before or after vaccination).
- The investigator or an authorized designee completes the CRF.

# 6.2.8. Group 2 Visit 8 (Prevnar 13: 12-Month Visit, 365 to 386 Days of Age)

- Ensure and document that the subject continues to be eligible for the study (see Section 6.5 for withdrawal information).
- Record vaccines administered since Visit 7 as described in Section 5.7.4.
- Determine whether any SAEs or NDCMCs have occurred since the previous visit and follow up on any previously reported events to determine the outcome (ie, record stop dates or confirm if they are still continuing) and record as described in Section 8, and record concomitant medications used to treat SAEs and NDCMCs.
- Administer a single 0.5-mL injection of Prevnar 13 into the right anterolateral thigh.

• Administer permitted vaccines (to be administered into a limb other than the left leg).

## After vaccination:

- Remind the subject's legally acceptable representative to contact the investigator or investigator site staff as soon as possible if any significant illness or medical event (eg, emergency room visit or hospitalization) occurs.
- Remind the subject's legally acceptable representative that use of prophylactic antipyretic/pain medication, while permitted, is not recommended on the day of investigational product administration (before or after vaccination).
- The investigator or an authorized designee completes the CRF and updates the investigational product accountability records.

# 6.2.9. Group 2 Visit 9 (c7vPnC Dose 4: 13-Month Visit, 21 to 35 Days After Prevnar 13 at Visit 8)

- Ensure and document that the subject continues to be eligible for the study (see Section 6.5 for withdrawal information), and none of the temporary delay criteria are met.
- Record vaccines administered since Visit 8 as described in Section 5.7.4.
- Determine whether any SAEs or NDCMCs have occurred since the previous visit and follow up on any previously reported events to determine the outcome (ie, record stop dates or confirm if they are still continuing) and record as described in Section 8, and record concomitant medications used to treat SAEs and NDCMCs.
- Measure and record the subject's rectal temperature (°F/°C).
- Collect a blood sample of approximately 5 mL for immunogenicity prior to vaccination (a topical anesthetic is permitted).
- Administer a single 0.5-mL injection of c7vPnC into the left anterolateral thigh.

- Site staff will observe the subject for at least 30 minutes after vaccination for any acute reactions. Record any AEs on the CRF and on an SAE form as applicable. Record concomitant medications used to treat SAEs and NDCMCs.
- Issue the subject's legally acceptable representative an e-diary (if device needed). Provide and review instructions on use and completion of the e-diary. Ask the subject's legally acceptable representative to complete the e-diary from Day 1 to Day 7, with Day 1 being the day of vaccination. Provide thermometer or measuring device if needed.

- Ask the subject's legally acceptable representative to contact the investigator site staff or investigator immediately during the 7-day postvaccination period if the subject experiences fever >104.0°F (>40.0°C), redness or swelling at the injection site measuring >14 measuring device units (>7 cm), or severe injection site pain (causes limitation of limb movement) to determine if the event requires further assessment by the investigator.
- Remind the subject's legally acceptable representative to contact the investigator or investigator site staff as soon as possible if any significant illness or medical event (eg, emergency room visit or hospitalization) occurs.
- Remind the subject's legally acceptable representative that use of prophylactic antipyretic/pain medication, while permitted, is not recommended on the day of investigational product administration (before or after vaccination).
- The investigator or an authorized designee completes the CRF and updates the investigational product accountability records.

## 6.2.10. Group 2 Visit 10 (Follow-up: 14-Month Visit, 28 to 42 Days After Dose 4)

- Ensure and document that the subject continues to be eligible for the study (see Section 6.5 for withdrawal information), and none of the temporary delay criteria are met.
- Record vaccines administered since Visit 9 as described in Section 5.7.4.
- Review the subject's e-diary data with the subject's legally acceptable representative; collect stop dates of any e-diary events ongoing on the last day that the e-diary was completed and record stop dates in the CRF.
- Collect the e-diary (if device provided).
- Determine whether any AEs (includes nonserious AEs, SAEs, or NDCMCs) have
  occurred since the previous visit and follow up on any previously reported events to
  determine the outcome (ie, record stop dates or confirm if they are still continuing) and
  record as described in Section 8, and record concomitant medications used to treat SAEs
  and NDCMCs.
- Collect a blood sample of approximately 5 mL for immunogenicity assessments (a topical anesthetic is permitted).
- Remind the subject's legally acceptable representative to contact the investigator or investigator site staff immediately if any significant illness or medical event (eg, emergency room visit or hospitalization) occurs.
- The investigator or an authorized designee completes the CRF.

# 6.2.11. Group 2 Visit 11 (Follow-up: 19-Month Phone Contact, 168 to 196 Days After Dose 4)

- Contact the subject's legally acceptable representative by telephone approximately 6 months after the last dose of c7vPnC; this contact should be attempted for all subjects who have received at least 1 dose of c7vPnC, unless the subject's legally acceptable representative has withdrawn consent.
- Determine whether any SAEs or NDCMCs have occurred since the previous visit and follow up on any previously reported events to determine the outcome (ie, record stop dates or confirm if they are still continuing) and record as described in Section 8, and record concomitant medications used to treat SAEs and NDCMCs.
- The investigator or an authorized designee completes the CRF.

# 6.3. Group 3 (Control With Supplemental Dose) Study Procedures

## 6.3.1. Group 3 Visit 1 (Dose 1: 2-Month Visit, Day 1)

Prior to randomization:

- A personally signed and dated informed consent document indicating that the subject's legally acceptable representative has been informed of all pertinent aspects of the study before performing any study-specific procedures.
- Record the subject's demographic information (including date of birth, sex, race, and ethnicity).
- Obtain and record the subject's medical history including prior vaccinations.
- Perform physical examination evaluating any clinically significant abnormalities within the following body systems: general appearance; skin; head, eyes, ears, nose, and throat; heart; lungs; abdomen; musculoskeletal; extremities; neurological; and lymph nodes. Clinically significant abnormal results will be recorded in the CRF.
- Measure and record the subject's rectal temperature (°F/°C).
- Ensure that all inclusion criteria, none of the exclusion criteria, and none of the temporary delay criteria are met.
- Assign randomization number and investigational container number via the IRT. This must be the last step before proceeding. A site staff member will prepare the investigational product according to the IP manual.

#### After randomization:

• Administer a single 0.5-mL injection of Prevnar 13 into the left anterolateral thigh.

- Administer DTaP-containing vaccine and other permitted vaccines (to be administered into a limb other than the site of Prevnar 13 injection).
- Site staff will observe the subject for at least 30 minutes after vaccination for any acute reactions. Record any AEs on the CRF and on an SAE form as applicable. Record concomitant medications used to treat SAEs and NDCMCs.
- Issue the subject's legally acceptable representative a measuring device to measure injection site reactions and a digital thermometer and provide instructions on their use.
- Issue the subject's legally acceptable representative an e-diary (device or application). Provide instructions on use and completion of the e-diary. Ask the subject's legally acceptable representative to complete the e-diary from Day 1 to Day 7, with Day 1 being the day of vaccination.
- Ask the subject's legally acceptable representative to contact the investigator or investigator site staff as soon as possible if any significant illness or medical event (eg, emergency room visit or hospitalization) occurs.
- Inform the subject's legally acceptable representative that use of prophylactic antipyretic/pain medication, while permitted, is not recommended on the day of investigational product administration (before or after vaccination).
- The investigator or an authorized designee completes the CRF and updates the investigational product accountability records.

## 6.3.2. Group 3 Visit 2 (Dose 2: 4-Month Visit, 42 to 63 Days After Dose 1)

- Ensure and document that the subject continues to be eligible for the study (see Section 6.5 for withdrawal information), and none of the temporary delay criteria are met.
- Record vaccines administered since Visit 1 as described in Section 5.7.4.
- Review the subject's e-diary data with the subject's legally acceptable representative; collect stop dates of any e-diary events ongoing on the last day that the e-diary was completed and record stop dates in the CRF.
- Determine whether any AEs (includes nonserious AEs, SAEs, and NDCMCs) have occurred since the previous visit and follow up on any previously reported events to determine the outcome (ie, record stop dates or confirm if they are still continuing) and record as described in Section 8, and record concomitant medications used to treat SAEs and NDCMCs.
- Measure and record the subject's rectal temperature ( ${}^{\circ}F/{}^{\circ}C$ ).
- Administer a single 0.5-mL injection of Prevnar 13 into the left anterolateral thigh.

• Administer DTaP-containing vaccine and other permitted vaccines (to be administered into a limb other than the site of Prevnar 13 injection).

#### After vaccination:

- Site staff will observe the subject for at least 30 minutes after vaccination for any acute reactions. Record any AEs on the CRF and on an SAE form as applicable. Record concomitant medications used to treat SAEs and NDCMCs.
- Confirm that the e-diary is working and review instructions if necessary. Remind the subject's legally acceptable representative to complete the e-diary from Day 1 to Day 7, with Day 1 being the day of vaccination. Provide thermometer or measuring device if needed.
- Remind the subject's legally acceptable representative to contact the investigator or investigator site staff as soon as possible if any significant illness or medical event (eg, emergency room visit or hospitalization) occurs during the study period.
- Remind the subject's legally acceptable representative that use of prophylactic antipyretic/pain medication, while permitted, is not recommended on the day of investigational product administration (before or after vaccination).
- The investigator or an authorized designee completes the CRF and updates the investigational product accountability records.

# 6.3.3. Group 3 Visit 3 (Dose 3: 6-Month Visit, 42 to 63 Days After Dose 2)

- Ensure and document that the subject continues to be eligible for the study (see Section 6.5 for withdrawal information), and none of the temporary delay criteria are met.
- Record vaccines administered since Visit 2 as described in Section 5.7.4.
- Review the subject's e-diary data with the subject's legally acceptable representative; collect stop dates of any e-diary events ongoing on the last day that the e-diary was completed and record stop dates in the CRF.
- Determine whether any AEs (includes nonserious AEs, SAEs, and NDCMCs) have
  occurred since the previous visit and follow up on any previously reported events to
  determine the outcome (ie, record stop dates or confirm if they are still continuing) and
  record as described in Section 8, and record concomitant medications used to treat SAEs
  and NDCMCs.
- Measure and record the subject's rectal temperature ( $^{\circ}F/^{\circ}C$ ).
- Administer a single 0.5-mL injection of Prevnar 13 into the left anterolateral thigh.

• Administer DTaP-containing vaccine and other permitted vaccines (to be administered into a limb other than the site of Prevnar 13 injection).

#### After vaccination:

- Site staff will observe the subject for at least 30 minutes after vaccination for any acute reactions. Record any AEs on the CRF and on an SAE form as applicable. Record concomitant medications used to treat SAEs and NDCMCs.
- Confirm that the e-diary is working and review instructions if necessary. Remind the subject's legally acceptable representative to complete the e-diary from Day 1 to Day 7, with Day 1 being the day of vaccination. Provide thermometer or measuring device if needed.
- Remind the subject's legally acceptable representative to contact the investigator or investigator site staff as soon as possible if any significant illness or medical event (eg, emergency room visit or hospitalization) occurs during the study period.
- Remind the subject's legally acceptable representative that use of prophylactic antipyretic/pain medication, while permitted, is not recommended on the day of investigational product administration (before or after vaccination).
- The investigator or an authorized designee completes the CRF and updates the investigational product accountability records.

# 6.3.4. Group 3 Visit 4 (Follow-up: 7-Month Visit, 28 to 42 Days After Dose 3)

- Ensure and document that the subject continues to be eligible for the study (see Section 6.5 for withdrawal information), and none of the temporary delay criteria are met.
- Record vaccines administered since Visit 3 as described in Section 5.7.4.
- Review the subject's e-diary data with the subject's legally acceptable representative; collect stop dates of any e-diary events ongoing on the last day that the e-diary was completed and record stop dates in the CRF.
- Collect the e-diary (if device provided).
- Determine whether any AEs (includes nonserious AEs, SAEs, and NDCMCs) have
  occurred since the previous visit and follow up on any previously reported events to
  determine the outcome (ie, record stop dates or confirm if they are still continuing) and
  record as described in Section 8, and record concomitant medications used to treat SAEs
  and NDCMCs.
- Collect a blood sample of approximately 5 mL for immunogenicity (a topical anesthetic is permitted).

- Remind the subject's legally acceptable representative to contact the investigator or investigator site staff as soon as possible if any significant illness or medical event (eg, emergency room visit or hospitalization) occurs during the study period.
- Inform the subject's legally acceptable representative that use of prophylactic antipyretic/pain medication, while permitted, is not recommended on the day of investigational product administration (before or after vaccination).
- The investigator or an authorized designee completes the CRF.

# 6.3.5. Group 3 Visit 5 (Dose 4: 12-Month Visit, 365 to 386 Days of Age)

- Ensure and document that the subject continues to be eligible for the study (see Section 6.5 for withdrawal information), and none of the temporary delay criteria are met.
- Record vaccines administered since Visit 4 as described in Section 5.7.4.
- Determine whether any SAEs or NDCMCs have occurred since the previous visit and follow up on any previously reported events to determine the outcome (ie, record stop dates or confirm if they are still continuing) and record as described in Section 8, and record concomitant medications used to treat SAEs and NDCMCs.
- Measure and record the subject's rectal temperature (°F/°C).
- Collect a blood sample of approximately 5 mL for immunogenicity prior to vaccination (a topical anesthetic is permitted).
- Administer a single 0.5-mL injection of Prevnar 13 into the left anterolateral thigh.
- Administer permitted vaccines (to be administered into a limb other than the site of Prevnar 13 injection).

- Site staff will observe the subject for at least 30 minutes after vaccination for any acute reactions. Record any AEs on the CRF and on an SAE form as applicable. Record concomitant medications used to treat SAEs and NDCMCs.
- Issue the subject's legally acceptable representative an e-diary (if device needed). Provide and review instructions on use and completion of the e-diary. Ask the subject's legally acceptable representative to complete the e-diary from Day 1 to Day 7, with Day 1 being the day of vaccination. Provide thermometer or measuring device if needed.
- Remind the subject's legally acceptable representative to contact the investigator or investigator site staff as soon as possible if any significant illness or medical event (eg, emergency room visit or hospitalization) occurs.

- Remind the subject's legally acceptable representative that use of prophylactic antipyretic/pain medication, while permitted, is not recommended on the day of investigational product administration (before or after vaccination).
- The investigator or an authorized designee completes the CRF and updates the investigational product accountability records.

# 6.3.6. Group 3 Visit 6 (Follow-up and Administration of the c7vPnC Supplemental Dose: 13-Month Visit, 28 to 42 Days After Dose 4)

- Ensure and document that the subject continues to be eligible for the study (see Section 6.5 for withdrawal information), and none of the temporary delay criteria are met.
- Record vaccines administered since Visit 5 as described in Section 5.7.4.
- Review the subject's e-diary data with the subject's legally acceptable representative; collect stop dates of any e-diary events ongoing on the last day that the e-diary was completed and record stop dates in the CRF.
- Determine whether any AEs (includes nonserious AEs, SAEs, or NDCMCs) have occurred since the previous visit and follow up on any previously reported events to determine the outcome (ie, record stop dates or confirm if they are still continuing) and record as described in Section 8, and record concomitant medications used to treat SAEs and NDCMCs.
- Measure and record the subject's rectal temperature (°F/°C).
- Collect a blood sample of approximately 5 mL for immunogenicity prior to vaccination (a topical anesthetic is permitted).
- Administer a single 0.5-mL injection of c7vPnC into the left anterolateral thigh.

- Site staff will observe the subject for at least 30 minutes after vaccination for any acute reactions. Record any AEs on the CRF and on an SAE form as applicable. Record concomitant medications used to treat SAEs and NDCMCs.
- Confirm that the e-diary is working and review instructions if necessary. Remind the subject's legally acceptable representative to complete the e-diary from Day 1 to Day 7, with Day 1 being the day of vaccination. Provide thermometer or measuring device if needed.
- Ask the subject's legally acceptable representative to contact the investigator site staff or investigator as soon as possible during the 7-day postvaccination period if the subject experiences fever >104.0°F (>40.0°C), redness or swelling at the injection site measuring

- >14 measuring device units (>7 cm), or severe injection site pain (causes limitation of limb movement) to determine if the event requires further assessment by the investigator.
- Remind the subject's legally acceptable representative to contact the investigator or investigator site staff immediately if any significant illness or medical event (eg, emergency room visit or hospitalization) occurs.
- Remind the subject's legally acceptable representative that use of prophylactic antipyretic/pain medication, while permitted, is not recommended on the day of investigational product administration (before or after vaccination).
- The investigator or an authorized designee completes the CRF and updates the investigational product accountability records.

# 6.3.7. Group 3 Visit 7 (Follow-up of the Supplemental Dose: 14-Month Visit, 28 to 42 Days After the Supplemental Dose)

- Ensure and document that the subject continues to be eligible for the study (see Section 6.5 for withdrawal information), and none of the temporary delay criteria are met.
- Record vaccines administered since Visit 6 as described in Section 5.7.4.
- Review the subject's e-diary data with the subject's legally acceptable representative; collect stop dates of any e-diary events ongoing on the last day that the e-diary was completed and record stop dates in the CRF.
- Collect the e-diary (if device provided).
- Determine whether any AEs (includes nonserious AEs, SAEs, or NDCMCs) have
  occurred since the previous visit and follow up on any previously reported events to
  determine the outcome (ie, record stop dates or confirm if they are still continuing) and
  record as described in Section 8, and record concomitant medications used to treat SAEs
  and NDCMCs.
- Remind the subject's legally acceptable representative to contact the investigator or investigator site staff immediately if any significant illness or medical event (eg, emergency room visit or hospitalization) occurs.
- The investigator or an authorized designee completes the CRF.

# 6.3.8. Group 3 Visit 8 (Follow-up: 19-Month Phone Contact, 168 to 196 Days After the Supplemental Dose)

- Contact the subject's legally acceptable representative by telephone approximately 6 months after the Supplemental Dose; this contact should be attempted for all subjects who have received at least 1 dose of Prevnar 13, unless the subject's legally acceptable representative has withdrawn consent.
- Determine whether any SAEs or NDCMCs have occurred since the previous visit and follow up on any previously reported events to determine the outcome (ie, record stop dates or confirm if they are still continuing) and record as described in Section 8, and record concomitant medications used to treat SAEs and NDCMCs.
- The investigator or an authorized designee completes the CRF.

## 6.4. Unscheduled Visits

If the subject's legally acceptable representative reports redness or swelling at the injection site measuring >14 measuring device units (>7 cm) or severe injection site pain or a fever >104.0°F (>40.0°C) during the 7-day postvaccination period of c7vPnC Doses 1 to 4 and the Supplemental Dose, a telephone contact must occur as soon as possible between the investigator or medically qualified designee and subject's legally acceptable representative to assess if an unscheduled investigator site visit is required. Note that for a fever >104.0°F (>40.0°C), the subject's legally acceptable representative should be instructed not to delay seeking medical care, as appropriate, while arranging for an unscheduled visit. An investigator site visit should be scheduled as soon as possible to assess the extent of the reaction unless any of the following is true:

- The subject's legally acceptable representative is unable to bring the subject to the unscheduled visit.
- The reaction is no longer present at the time of the telephone contact.
- The subject's legally acceptable representative recorded an incorrect value in the e-diary (confirmation of an e-diary data entry error).
- The principal investigator (PI) or authorized designee determined it was not needed.

This telephone contact will be recorded in the subject's source documentation and the CRF.

If the subject's legally acceptable representative is unable to bring the subject to an unscheduled visit, or the PI or authorized designee determined it was not needed, any ongoing reactions must be assessed at the next study visit.

During the investigator site visit, the reactions should be assessed by the investigator or a medically qualified member of the study staff such as a study physician or a study nurse, as applicable to the investigator's local practice, who will:

- Measure rectal temperature (°F/°C).
- Measure minimum and maximum diameters of redness (if present).
- Measure minimum and maximum diameters of swelling (if present).
- Assess injection site pain in accordance with the grades provided in Section 7.1.2 (if present).
- Assess for other findings associated with the reaction and record on the AE page of the CRF, if appropriate.

The investigator or an authorized designee will complete the unscheduled visit assessment page of the CRF.

The subject's legally acceptable representative will also be instructed to contact investigator site staff if the subject experiences any emergency room visit or hospitalization for decreased appetite, drowsiness/increased sleep, irritability, or local reaction within 7 days of vaccination.

The subject's legally acceptable representative will also be instructed to contact the investigator site to report any significant illness, medical event, or hospitalization that occurs during the study period. The investigator site should determine if an unscheduled visit to further evaluate the event is warranted in all such cases.

Additionally, study staff may contact the subject's legally acceptable representative to obtain additional information on Grade 3 events entered into the e-diary.

## 6.5. Subject Withdrawal

An investigator and/or sponsor can withdraw a subject from the study if deemed appropriate. In addition, if a subject fails to continue to meet applicable inclusion criteria, new information becomes available that would exclude the subject, or the subject develops a condition or situation that would meet exclusion criteria (eg, exclusion criteria 1, 6 to 13), the subject may be considered for withdrawal.

Reasons why a subject may discontinue or be withdrawn from the study by the investigator or sponsor include, but are not limited to, failure to meet entrance criteria (screening failure), AE, death, protocol deviation, lost to follow-up, legally acceptable representative no longer willing to participate in the study, study terminated by the sponsor, or any other reason. Subjects who have received the investigational product will not be replaced regardless of the reason for withdrawal.

The investigator should capture the reason for withdrawal in the database for all subjects and a follow-up telephone contact for the collection of safety information should be completed for all subjects who have been withdrawn after administration of investigational product unless consent for further contact has been withdrawn.

The subject's legally acceptable representative may withdraw the study subject from the study at any time at the representative's own request, or the subject may be withdrawn at any time at the discretion of the investigator or sponsor for safety (see also the Withdrawal From the Study Due to Adverse Events, Section 8.1.3) or behavioral reasons, or the inability of the subject or the subject's legally acceptable representative to comply with the protocol-required schedule of study visits or procedures at a given study site.

If a subject does not return for a scheduled visit, every effort should be made to contact the subject's legally acceptable representative. All attempts to contact the subject's legally acceptable representative and information received during contact attempts must be documented in the subject's medical record. In any circumstance, every effort should be made to document subject outcome, if possible. The investigator should inquire about the reason for withdrawal, request that the subject return for a final visit, if applicable, and follow up with the subject regarding any unresolved AEs.

If the subject's legally acceptable representative withdraws the subject from the study, and also withdraws consent for disclosure of future information, no further evaluations should be performed, and no additional data should be collected. The sponsor may retain and continue to use any data collected before such withdrawal of consent.

#### Withdrawal of consent:

Subjects whose legally acceptable representative requests the subject to discontinue receipt of investigational product will remain in the study and must continue to be followed for protocol-specified safety procedures through 6 months after the last dose of c7vPnC for Groups 1 and 2 and the c7vPnC Supplemental Dose for Group 3. The only exception to this is when the subject's legally acceptable representative specifically withdraws consent for any further contact with the subject. The subject's legally acceptable representative should notify the investigator in writing of the decision to withdraw consent from future follow-up, whenever possible. The withdrawal of consent should be explained in detail in the medical records by the investigator, as to whether the withdrawal is only from further receipt of investigational product or also from study procedures and/or posttreatment study follow-up, and entered on the appropriate CRF page.

#### Lost to follow-up:

All reasonable efforts must be made to locate the subject and/or the subject's legally acceptable representative to determine and report their ongoing status. This includes follow-up with persons authorized by the subject as noted above. Lost to follow-up is defined by the inability to reach the subject's legally acceptable representative after a minimum of 2 documented phone calls, faxes, or emails as well as lack of response by the subject's legally acceptable representative to 1 registered mail letter. All attempts should be documented in the subject's medical records. If it is determined that the subject has died, the site will use locally permissible methods to obtain the date and cause of death. If the investigator's use of a third-party representative to assist in the follow-up portion of the study has been included in the subject's informed consent, then the investigator may use a

Final Protocol Amendment 1, 18 Feb 2020

sponsor-retained third-party representative to assist site staff with obtaining the subject's contact information or other public vital status data necessary to complete the follow-up portion of the study. The site staff and representative will consult publicly available sources, such as public health registries and databases, in order to obtain updated contact information. If, after all attempts, the subject remains lost to follow-up, then the last-known-alive date as determined by the investigator should be reported and documented in the subject's medical records.

### 7. ASSESSMENTS

Every effort should be made to ensure that the protocol-required tests and procedures are completed as described. However, it is anticipated that from time to time there may be circumstances outside of the control of the investigator that may make it unfeasible to perform the test. In these cases the investigator will take all steps necessary to ensure the safety and well-being of the subject. When a protocol-required test cannot be performed, the investigator will document the reason for this and any corrective and preventive actions that he or she has taken to ensure that normal processes are adhered to as soon as possible. The study team will be informed of these incidents in a timely manner.

## 7.1. Safety Parameters

Safety parameters will be assessed as described in the Schedule of Activities, Section 8, and below.

A medical history, physical examination, and measurement of rectal temperature will be performed on all subjects prior to Dose 1 of c7vPnC in Groups 1 and 2 and the first dose of Prevnar 13 in Group 3 to determine subject eligibility and to establish a clinical baseline. Significant medical history and clinically significant observations from the physical examination and temperature measurement will be documented and recorded in the CRF.

Acute reactions within the first 30 minutes after Doses 1 to 4, the c7vPnC Supplemental Dose (Group 3), and concomitant vaccine administration (Groups 1 and 3) will be assessed and documented as an AE or SAE in the CRF, as appropriate. Prompted e-diary events, including local reactions (pain, redness, and swelling) and systemic events (fever, decreased appetite, drowsiness/increased sleep, and irritability) that occur in the 7 days after Doses 1 to 4 and the Supplemental Dose, are graded as described in Section 7.1.2.

# 7.1.1. Subject Electronic Diary

The subject's legally acceptable representative will be asked to monitor and record local reactions, specific systemic events, and antipyretic/pain medication taken for 7 days, each evening following Doses 1 to 4 and the Supplemental Dose using an e-diary (in a provisioned device or an application on a personal device), which allows recording of these assessments only within a fixed time window, thus providing the accurate representation of the subject's experience at that time. Data on local reactions, specific systemic events, and antipyretic/pain medication reported in the e-diary will be transferred electronically to the e-diary vendor, where they will be available for review by investigators, their qualified designees, and sponsor staff at all times via an internet-based portal. At intervals agreed to

by the vendor and Pfizer, these data will be transferred electronically to Pfizer for analysis and reporting.

The daily e-diary data will not be captured in the CRF. However, if a subject withdraws because of prompted events reported in the e-diary, the event(s) should be recorded on the AE page of the CRF, regardless of whether the investigator considers the event(s) to be clinically significant.

The investigator or designee must obtain stop dates for any reactions ongoing on the last day that the e-diary was completed. The stop dates should be entered in the CRF.

Investigators (or an appropriately qualified designee) are required to review the e-diary data online at frequent intervals (daily is optimal) to evaluate subject compliance and reported events as part of the ongoing safety review.

# 7.1.2. Grading Scale for Prompted Events

The grading scales used in this study to assess prompted events as described below are based on concepts outlined in the Food and Drug Administration (FDA) Center for Biologics Evaluation and Research (CBER) guidelines on toxicity grading scales for adults and adolescent volunteers enrolled in preventive vaccine clinical trials, but have been adapted for applicability to healthy infants.<sup>69</sup>

#### 7.1.2.1. Local Reactions

For the first 7 days following Doses 1 to 4 and the Supplemental Dose, the subject's legally acceptable representative will be asked to assess redness, swelling, and pain at the injection site and to record the symptoms in the e-diary in the evening. Redness and swelling will be measured and recorded in measuring device units (range: 1 to >14; an entry in the e-diary of 15 will denote >14), and then categorized during analysis as mild, moderate, or severe based on the grading scale in Table 2 below. Measuring device units can be converted to centimeters according to the following scale: 1 measuring device unit = 0.5 cm. Pain at the vaccine injection site will be assessed by the subject's legally acceptable representative as mild, moderate, or severe according to the grading scale in Table 2 below. The subject's legally acceptable representative will be prompted to contact the investigator if the subject experiences a severe (Grade 3 or above) local reaction to assess the reaction and perform an unscheduled assessment or visit as appropriate.

Only an investigator is able to classify a subject's local reaction as Grade 4, after physical examination of the subject or documentation from another medically qualified source (eg, emergency room or hospital record). If a subject experiences a Grade 4 local reaction, the investigator must immediately notify the sponsor. Site staff will educate the subject's legally acceptable representative regarding signs and symptoms that would prompt site contact.

The procedure for notification of the sponsor is provided in the study reference manual (SRM) or equivalent.

**Table 2.** Grading Scales for Local Reactions

| | Mild<br>Grade 1 | Moderate<br>Grade 2 | Severe<br>Grade 3 <sup>a</sup> | Grade 4 <sup>b</sup> |
|---|---|---|---|---|
| Redness<br>(synonymous with<br>erythema) | 1 to 4 caliper units (or<br>measuring device<br>units)<br>=<br>0.5 to 2.0 cm | 5 to 14 caliper units (or<br>measuring device<br>units)<br>=<br>>2.0 to 7.0 cm | >14 caliper units (or<br>measuring device<br>units)<br>=<br>>7 cm | Necrosis or exfoliative dermatitis |
| Swelling<br>(synonymous with<br>edema) | 1 to 4 caliper units (or measuring device units) = 0.5 to 2.0 cm | 5 to 14 caliper units (or measuring device units) = >2.0 to 7.0 cm | >14 caliper units (or<br>measuring device<br>units)<br>=<br>>7 cm | Necrosis |
| Pain at injection site (tenderness) | Hurts if gently touched<br>(eg, whimpers, winces,<br>protests, or withdraws) | Hurts if gently touched, with crying | Causes limitation of limb movement | Emergency room visit<br>or hospitalization for<br>severe pain<br>(tenderness) at<br>injection site |

Abbreviations: CRF = case report form; e-diary = electronic diary.

Note: If the size of the redness and/or swelling falls between 2 measuring device units, the higher measuring device unit number will be recorded in the e-diary.

- a. Legally acceptable representatives of the subjects experiencing local reactions >14 caliper units (>7.0 cm) are to be contacted by the study site. An unscheduled visit may be required.
- b. Grade 4 assessment should be made by the investigator. Grade 4 will not be collected in the e-diary but as an AE on the CRF. The severity of the local reaction should be graded using the AE severity grading scale in Section 8.3.

# 7.1.2.2. Systemic Event Symptoms and Fever

## 7.1.2.2.1. Systemic Event Symptoms

For the first 7 days following Doses 1 to 4 and the Supplemental Dose, the subject's legally acceptable representative will be asked to assess decreased appetite, drowsiness/increased sleep, and irritability and to record the symptoms in the e-diary in the evening. The symptoms will be assessed by the subject's legally acceptable representative as mild, moderate, or severe according to the grading scale in Table 3 below. The subject's legally acceptable representative will also be instructed to contact site staff if the subject experiences any possible Grade 4 prompted systemic event (ie, emergency room visit or hospitalization for severe decreased appetite, severe drowsiness/increased sleep, or severe irritability) within 7 days after vaccination. Study staff may also contact the subject's legally acceptable representative to obtain additional information on Grade 3 events entered into the e-diary.

Only an investigator is able to classify a subject's systemic event as Grade 4, after physical examination of the subject or documentation from another medically qualified source (eg, emergency room or hospital record) or telephone contact with the subject's legally acceptable representative. If a subject experiences a Grade 4 systemic event, the investigator must immediately notify the sponsor.

The procedure for notification of the sponsor is provided in the SRM or equivalent.

**Table 3.** Grading Scales for Systemic Events

| Systemic Event | Mild | Moderate | Severe | |
|---|---|---|---|---|
| - | Grade 1 | Grade 2 | Grade 3 | Grade 4 <sup>a</sup> |
| Decreased appetite | Decreased interest in | Decreased oral | Refusal to feed | Emergency room |
| (loss of appetite) | eating | intake | | visit or |
| | | | | hospitalization for |
| | | | | severe decreased |
| | | | | appetite (loss of |
| | | | | appetite) |
| Drowsiness | Increased or | Slightly subdued, | Disabling, not | Emergency room |
| (increased sleep) | prolonged sleeping | interfering with daily | interested in usual | visit or |
| | bouts | activity | daily activity | hospitalization for |
| | | | | severe drowsiness |
| | | | | (increased sleep) |
| Irritability | Easily consolable | Requiring increased | Inconsolable; crying | Emergency room |
| (fussiness) | | attention | cannot be comforted | visit or |
| | | | | hospitalization for |
| (synonymous with | | | | severe irritability |
| restless sleep; | | | | (fussiness) |
| decreased sleep) | | | | |

Abbreviations: CRF = case report form; e-diary = electronic diary.

## 7.1.2.2.2. Fever

In order to record information on fever, a digital thermometer will be given to the subject's legally acceptable representative with instructions on how to measure rectal temperature at home. Temperature will be collected in the evening daily for 7 days following Doses 1 to 4 and the Supplemental Dose (Days 1 to 7, where Day 1 is the day of vaccination) and at any time during the 7 days that fever is suspected. Fever is defined as a rectal temperature of  $\geq 100.4^{\circ}F$  ( $\geq 38.0^{\circ}C$ ). The highest temperature for each day will be recorded in the e-diary. In the event of a fever on Day 7, temperature will be collected daily until fever has resolved (1 day of temperature less than  $100.4^{\circ}F$  [ $38.0^{\circ}C$ ]) in order to collect a stop date in the CRF. A subject's legally acceptable representative will be prompted to contact the investigator if the subject experiences a fever  $\geq 104.0^{\circ}F$  ( $\geq 40.0^{\circ}C$ ) to assess the fever and perform an unscheduled assessment. Study staff may also contact the subject's legally acceptable representative to obtain additional information if a temperature of  $\geq 102^{\circ}F$  is entered into an e-diary. Temperature will be measured and recorded to 1 decimal place and then grouped into ranges for the analysis; see Table 4 below.

a. Grade 4 assessment should be made by the investigator; Grade 4 will not be collected in the e-diary but will be collected as an AE on the CRF. The severity of the systemic event should be graded using the AE severity grading scale in Section 8.3.

# **Table 4.** Ranges for Fever

| 100.4°F to 101.1°F (38.0°C to 38.4°C) |
|---------------------------------------|
| 101.2°F to 102.0°F (38.5°C to 38.9°C) |
| 102.1°F to 104.0°F (39.0°C to 40.0°C) |
| >104.0°F (>40.0°C) |



# 7.2. Immunogenicity

Blood samples (approximately 5 mL/visit) for immunogenicity assessments will be collected from all subjects 1 month after Dose 3, prior to Dose 4, and 1 month after Dose 4, CCI.

In Group 2, blood will also be collected prior to Dose 3. Sample collection, processing, storage, and shipping information can be found in the SRM or equivalent manual.

Concentrations of anticapsular polysaccharide IgG antibodies for the 7 vaccine serotypes will be determined on sera collected at each blood draw in all subjects. The serotype-specific IgG concentrations will be measured by Pfizer's Luminex-based assay.



For samples being collected and shipped, detailed collection, processing, storage, and shipment instructions and contact information will be provided to the investigator site prior to initiation of the study. Serum samples should be processed and stored as indicated in the SRM or equivalent document.

Immunogenicity assays will be performed at the Pfizer Vaccine Research & Development laboratory located at 401 North Middletown Road, Pearl River, New York 10965 and/or at an external laboratory designated by Pfizer.

# 7.3. Biological Samples

Blood samples will be used only for scientific research. Each sample will be labeled with a code so that the laboratory personnel testing the samples will not know the subject's identity.

Samples that remain after performing assays outlined in the protocol may be stored by Pfizer. Unless a time limitation is required by local regulations or ethical requirements, the samples will be stored for up to 15 years after the end of the study and then destroyed.

No testing of the subject's genetic material will be performed.

The subject's legally acceptable representative may request that his or her child's samples, if still identifiable, be destroyed at any time; however, any data already collected from those samples will still be used for this research. The biological samples may be shared with other researchers as long as confidentiality is maintained and no testing of the subject's genetic material is performed.







## 8. ADVERSE EVENT REPORTING

## 8.1. Requirements

The table below summarizes the requirements for recording safety events on the CRF and for reporting safety events on the Clinical Trial (CT) SAE Report Form to Pfizer Safety. These requirements are delineated for 3 types of events: (1) SAEs; (2) nonserious AEs; and (3) exposure to the investigational product under study during pregnancy or breastfeeding, and occupational exposure.

| Safety Event | Recorded on the CRF | Reported on the CT SAE<br>Report Form to Pfizer |
|---|---|---|
| | | Safety Within 24 Hours of |
| | | Awareness |
| SAE | All | All |
| Nonserious AE <sup>a</sup> | All | None |
| Exposure to the | All (regardless of whether | Exposure during pregnancy, |
| investigational product | associated with an AE), except | exposure via breastfeeding, |
| under study during | occupational exposure | occupational exposure |
| pregnancy or breastfeeding, | | (regardless of whether |
| and occupational exposure | | associated with an AE) |

a. Nonserious AEs will be recorded from the time the subject provides informed consent through 1 month after Dose 3 and from Dose 4 to 1 month after Dose 4/Supplemental Dose. Newly diagnosed chronic medical conditions (can be nonserious) and SAEs will be reported from the time the subject provides informed consent through 6 months after Dose 4/Supplemental Dose.

All observed or volunteered events regardless of vaccine group or suspected causal relationship to the investigational product(s) will be reported as described in the following paragraphs.

Events listed in the table above that require reporting to Pfizer Safety on the CT SAE Report Form within 24 hours of awareness of the event by the investigator are to be reported regardless of whether the event is determined by the investigator to be related to an investigational product under study. In particular, if the SAE is fatal or life-threatening, notification to Pfizer Safety must be made immediately, irrespective of the extent of available event information. This time frame also applies to additional new (follow-up) information on previously forwarded reports. In the rare situation that the investigator does not become immediately aware of the occurrence of an event, the investigator must report the event within 24 hours after learning of it and document the time of his/her first awareness of the event.

For each event, the investigator must pursue and obtain adequate information both to determine the outcome and to assess whether it meets the criteria for classification as an SAE

Final Protocol Amendment 1, 18 Feb 2020

(see the SAE section below). In addition, the investigator may be requested by Pfizer Safety to obtain specific follow-up information in an expedited fashion. This information is more detailed than that recorded on the CRF. In general, this will include a description of the event in sufficient detail to allow for a complete medical assessment of the case and independent determination of possible causality. Any information relevant to the event, such as concomitant medications and illnesses, must be provided. In the case of a subject death, a summary of available autopsy findings must be submitted as soon as possible to Pfizer Safety. Any pertinent additional information must be reported on the CT SAE Report Form; additional source documents (eg, medical records, CRF, laboratory data) are to be sent to Pfizer Safety **ONLY** upon request.

As part of ongoing safety reviews conducted by the sponsor, any nonserious AE that is determined by the sponsor to be serious will be reported by the sponsor as an SAE. To assist in the determination of case seriousness, further information may be requested from the investigator to provide clarity and understanding of the event in the context of the clinical study.

## 8.1.1. Additional Details on Recording Adverse Events on the CRF

All events detailed in the table above will be recorded on the AE page(s) of the CRF. It should be noted that the CT SAE Report Form for reporting of SAE information is not the same as the AE page of the CRF. When the same data are collected, the forms must be completed in a consistent manner. AEs should be recorded using concise medical terminology and the same AE term should be used on both the CRF and the CT SAE Report Form for reporting of SAE information.

## 8.1.2. Eliciting Adverse Event Information

The investigator is to record on the CRF all directly observed AEs and all AEs spontaneously reported by the study subject's legally acceptable representative. In addition, each study subject's legally acceptable representative will be questioned about the occurrence of AEs in a nonleading manner.

# 8.1.3. Withdrawal From the Study Due to Adverse Events (see also the Subject Withdrawal Section)

Withdrawal due to AEs should be distinguished from withdrawal due to other causes, according to the definition of AE noted below, and recorded on the CRF.

When a subject withdraws from the study because of an SAE, the SAE must be recorded on the CRF and reported, as appropriate, on the CT SAE Report Form, in accordance with the Requirements section above.

## 8.1.4. Time Period for Collecting AE/SAE/NDCMC Information

The time period for actively eliciting and collecting AEs, SAEs, and NDCMCs ("active collection period") for each subject begins from the time the subject's legally acceptable representative provides informed consent, which is obtained before the subject's participation in the study (ie, before undergoing any study-related procedure and/or receiving

investigational product). AEs will be collected through 1 month after Dose 3 and from Dose 4 through 1 month after Dose 4 or 1 month after the Supplemental Dose in Group 3. NDCMCs and SAEs will be collected from signing of informed consent through 6 months after Dose 4 or the Supplemental Dose. An NDCMC is defined as a disease or medical condition, not previously identified, that is expected to be persistent or is otherwise long-lasting in its effects.

For subjects who are screen failures, the active collection period ends when screen failure status is determined.

# 8.1.4.1. Reporting SAEs to Pfizer Safety

All SAEs occurring in a subject during the active collection period are reported to Pfizer Safety on the CT SAE Report Form.

SAEs occurring in a subject after the active collection period has ended are reported to Pfizer Safety if the investigator becomes aware of them; at a minimum, all SAEs that the investigator believes have at least a reasonable possibility of being related to investigational product must be reported to Pfizer Safety.

Follow-up by the investigator continues throughout and after the active collection period and until the event or its sequelae resolve or stabilize at a level acceptable to the investigator, and Pfizer concurs with that assessment.

## 8.1.4.2. Recording Nonserious AEs and SAEs on the CRF

During the active collection period, both nonserious AEs and SAEs are recorded on the CRF.

Follow-up by the investigator may be required until the event or its sequelae resolve or stabilize at a level acceptable to the investigator, and Pfizer concurs with that assessment.

# 8.1.5. Causality Assessment

The investigator's assessment of causality must be provided for all AEs (serious and nonserious); the investigator must record the causal relationship on the CRF, and report such an assessment in accordance with the SAE reporting requirements, if applicable. An investigator's causality assessment is the determination of whether there exists a reasonable possibility that the investigational product caused or contributed to an AE; generally the facts (evidence) or arguments to suggest a causal relationship should be provided. If the investigator does not know whether or not the investigational product caused the event, then the event will be handled as "related to investigational product" for reporting purposes, as defined by the sponsor. If the investigator's causality assessment is "unknown but not related" to investigational product, this should be clearly documented on study records.

In addition, if the investigator determines that an SAE is associated with study procedures, the investigator must record this causal relationship in the source documents and CRF, and report such an assessment in the dedicated section of the CT SAE Report Form and in accordance with the SAE reporting requirements.

## 8.1.6. Sponsor's Reporting Requirements to Regulatory Authorities

AE reporting, including suspected unexpected serious adverse reactions, will be carried out in accordance with applicable local regulations.

#### 8.2. Definitions

#### 8.2.1. Adverse Events

An AE is any untoward medical occurrence in a study subject administered a product or medical device; the event need not necessarily have a causal relationship with the treatment or usage. Examples of AEs include, but are not limited to:

- Abnormal test findings;
- Clinically significant signs and symptoms;
- Changes in physical examination findings;
- Hypersensitivity;
- Progression/worsening of underlying disease;
- Drug abuse;
- Drug dependency.

Additionally, AEs may include signs and symptoms resulting from:

- Drug overdose;
- Drug withdrawal;
- Drug misuse;
- Drug interactions;
- Extravasation;
- Exposure during pregnancy (EDP);
- Exposure via breastfeeding;
- Medication error;
- Occupational exposure.

Events that, in the clinical judgment of the investigator, are 1) consistent with normal growth and development and 2) do not differ significantly in frequency or severity from expected,

are not generally to be considered AEs. Examples may include, but are not limited to, teething, contact diaper rash, spitting up, colic, or typical fussiness/crying in infants and children.

## 8.2.2. Abnormal Test Findings

Abnormal objective test findings should be recorded as AEs when any of the following conditions are met:

- Test result is associated with accompanying symptoms; and/or
- Test result requires additional diagnostic testing or medical/surgical intervention; and/or
- Test result leads to a change in study dosing (outside of any protocol-specified dose adjustments) or discontinuation from the study, significant additional concomitant drug treatment, or other therapy; and/or
- Test result is considered to be an AE by the investigator or sponsor.

Merely repeating an abnormal test, in the absence of any of the above conditions, does not constitute an AE. Any abnormal test result that is determined to be an error does not require recording as an AE.

## 8.2.3. Serious Adverse Events

A serious adverse event is any untoward medical occurrence at any dose that:

- Results in death;
- Is life-threatening (immediate risk of death);
- Requires inpatient hospitalization or prolongation of existing hospitalization;
- Results in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions);
- Results in congenital anomaly/birth defect.

Or that is considered to be:

• An important medical event.

Medical and scientific judgment is exercised in determining whether an event is an important medical event. An important medical event may not be immediately life-threatening and/or result in death or hospitalization. However, if it is determined that the event may jeopardize the subject or may require intervention to prevent one of the other AE outcomes, the important medical event should be reported as serious.

Examples of such events are intensive treatment in an emergency room or at home for allergic bronchospasm; blood dyscrasias or convulsions that do not result in hospitalization; or development of drug dependency or drug abuse.

Medical device complaints may meet the SAE reporting requirement criteria (see the Medical Device Complaint Reporting Requirements section). An incident is any malfunction (ie, the failure of a device to meet its performance specifications or to perform as intended; performance specifications include all claims made in the labeling for the device) that, directly or indirectly, might lead to or might have led to the death of a subject, or user, or of other persons, or to a serious deterioration in their state of health.

A serious injury that can cause a serious deterioration in state of health can include:

- A life-threatening illness, even if temporary in nature;
- A permanent impairment of a body function or permanent damage to a body structure;
- A condition necessitating medical or surgical intervention to prevent the above 2 bulleted items;

Examples: clinically relevant increase in the duration of a surgical procedure; a condition that requires hospitalization or significant prolongation of existing hospitalization;

- Any indirect harm as a consequence of an incorrect diagnostic or in vitro diagnostic device test results when used within the manufacturer's instructions for use;
- Fetal distress, fetal death, or any congenital abnormality or birth defects.

## 8.2.4. Hospitalization

Hospitalization is defined as any initial admission (even less than 24 hours) in a hospital or equivalent healthcare facility, or any prolongation of an existing admission. Admission also includes transfer within the hospital to an acute/intensive care unit (eg, from the psychiatric wing to a medical floor, medical floor to a coronary care unit, or neurological floor to a tuberculosis unit). An emergency room visit does not necessarily constitute a hospitalization; however, the event leading to the emergency room visit is assessed for medical importance.

Hospitalization does not include the following:

- Rehabilitation facilities;
- Hospice facilities;
- Respite care (eg, caregiver relief);
- Skilled nursing facilities;
- Nursing homes;
- Same-day surgeries (as outpatient/same-day/ambulatory procedures).

Hospitalization or prolongation of hospitalization in the absence of a precipitating clinical AE is not in itself an SAE. Examples include:

- Admission for treatment of a preexisting condition not associated with the development of a new AE or with a worsening of the preexisting condition (eg, for workup of a persistent pretreatment laboratory abnormality);
- Social admission (eg, subject has no place to sleep);
- Administrative admission (eg, for yearly physical examination);
- Protocol-specified admission during a study (eg, for a procedure required by the study protocol);
- Optional admission not associated with a precipitating clinical AE (eg, for elective cosmetic surgery);
- Hospitalization for observation without a medical AE;
- Preplanned treatments or surgical procedures. These should be noted in the baseline documentation for the entire protocol and/or for the individual subject.

Diagnostic and therapeutic noninvasive and invasive procedures, such as surgery, should not be reported as SAEs. However, the medical condition for which the procedure was performed should be reported if it meets the definition of an SAE. For example, an acute appendicitis that begins during the reporting period should be reported if the SAE requirements are met, and the resulting appendectomy should be recorded as treatment of the AE.

# 8.3. Severity Assessment

| GRADE | If required on the AE page of the CRF, the investigator will use the adjectives MILD, MODERATE, or SEVERE to describe the maximum intensity of the AE. For purposes of consistency, these intensity grades are defined as follows: | |
|---|---|---|
| 1 | MILD | Does not interfere with subject's usual function. |
| 2 | MODERATE | Interferes to some extent with subject's usual function. |
| 3 | SEVERE | Interferes significantly with subject's usual function. |

Note the distinction between the severity and the seriousness of an AE. A severe event is not necessarily an SAE. For example, a headache may be severe (interferes significantly with the subject's usual function) but would not be classified as serious unless it met one of the criteria for SAEs, listed above.

#### **8.4. Special Situations**

# 8.4.1. Protocol-Specified Serious Adverse Events

There are no protocol-specified SAEs in this study. All SAEs will be reported to Pfizer Safety by the investigator as described in previous sections, and will be handled as SAEs in the safety database.

# 8.4.2. Potential Cases of Drug-Induced Liver Injury

Humans exposed to a drug who show no sign of liver injury (as determined by elevations in transaminases) are termed "tolerators," while those who show transient liver injury, but adapt are termed "adaptors." In some subjects, transaminase elevations are a harbinger of a more serious potential outcome. These subjects fail to adapt and therefore are "susceptible" to progressive and serious liver injury, commonly referred to as drug-induced liver injury (DILI). Subjects who experience a transaminase elevation above 3 times the upper limit of normal (× ULN) should be monitored more frequently to determine if they are an "adaptor" or are "susceptible."

Liver function tests (LFTs) are not required as a routine safety monitoring procedure in this study. However, should an investigator deem it necessary to assess LFTs because a subject presents with clinical signs/symptoms, such LFT results should be managed and followed as described below.

In the majority of DILI cases, elevations in aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) precede total bilirubin (TBili) elevations (>2 × ULN) by several days or weeks. The increase in TBili typically occurs while AST/ALT is/are still elevated above 3 × ULN (ie, AST/ALT and TBili values will be elevated within the same laboratory sample). In rare instances, by the time TBili elevations are detected, AST/ALT values might have decreased. This occurrence is still regarded as a potential DILI. Therefore, abnormal elevations in either AST OR ALT in addition to TBili that meet the criteria outlined below are considered potential DILI (assessed per Hy's law criteria) cases and should always be considered important medical events, even before all other possible causes of liver injury have been excluded.

The threshold of laboratory abnormalities for a potential DILI case depends on the subject's individual baseline values and underlying conditions. Subjects who present with the following laboratory abnormalities should be evaluated further as potential DILI (Hy's law) cases to definitively determine the etiology of the abnormal laboratory values:

• Subjects with AST/ALT and TBili baseline values within the normal range who subsequently present with AST OR ALT values >3 × ULN AND a TBili value

- >2 × ULN with no evidence of hemolysis and an alkaline phosphatase value <2 × ULN or not available;
- For subjects with baseline AST **OR** ALT **OR** TBili values above the ULN, the following threshold values are used in the definition mentioned above, as needed, depending on which values are above the ULN at baseline:
  - Preexisting AST or ALT baseline values above the normal range: AST or ALT values >2 times the baseline values AND >3 × ULN; or >8 × ULN (whichever is smaller).
  - Preexisting values of TBili above the normal range: TBili level increased from baseline value by an amount of at least 1 × ULN or if the value reaches >3 × ULN (whichever is smaller).

Rises in AST/ALT and TBili separated by more than a few weeks should be assessed individually based on clinical judgment; any case where uncertainty remains as to whether it represents a potential Hy's law case should be reviewed with the sponsor.

The subject should return to the investigator site and be evaluated as soon as possible, preferably within 48 hours from awareness of the abnormal results. This evaluation should include laboratory tests, detailed history, and physical assessment.

In addition to repeating measurements of AST and ALT and TBili, laboratory tests should include albumin, creatine kinase (CK), direct and indirect bilirubin, gamma-glutamyl transferase (GGT), prothrombin time (PT)/international normalized ratio (INR), total bile acids, alkaline phosphatase, and acetaminophen drug and/or protein adduct levels. Consideration should also be given to drawing a separate tube of clotted blood and an anticoagulated tube of blood for further testing, as needed, for further contemporaneous analyses at the time of the recognized initial abnormalities to determine etiology. A detailed history, including relevant information, such as review of ethanol, acetaminophen (either by itself or as a coformulated product in prescription or over-the-counter medications), recreational drug, supplement (herbal) use and consumption, family history, sexual history, travel history, history of contact with a jaundiced person, surgery, blood transfusion, history of liver or allergic disease, and potential occupational exposure to chemicals, should be collected. Further testing for acute hepatitis A, B, C, D, and E infection and liver imaging (eg, biliary tract) may be warranted.

All cases demonstrated on repeat testing as meeting the laboratory criteria of AST/ALT and TBili elevation defined above should be considered potential DILI (Hy's law) cases if no other reason for the LFT abnormalities has yet been found. Such potential DILI (Hy's law) cases are to be reported as SAEs, irrespective of availability of all the results of the investigations performed to determine etiology of the LFT abnormalities.

A potential DILI (Hy's law) case becomes a confirmed case only after all results of reasonable investigations have been received and have excluded an alternative etiology.

# 8.4.3. Exposure to the Investigational Product During Pregnancy or Breastfeeding, and Occupational Exposure

Exposure to the investigational product under study during pregnancy or breastfeeding and occupational exposure are reportable to Pfizer Safety within 24 hours of investigator awareness.

# **8.4.3.1.** Exposure During Pregnancy

For both unapproved/unlicensed products and for marketed products, an exposure during pregnancy (EDP) occurs if:

- A female becomes, or is found to be, pregnant either while receiving or having been exposed (eg, because of treatment or environmental exposure) to the investigational product; or the female becomes or is found to be pregnant after discontinuing and/or being exposed to the investigational product;
  - An example of environmental exposure would be a case involving direct contact with a Pfizer product in a pregnant woman (eg, a nurse reports that she is pregnant and has been exposed to chemotherapeutic products).
- A male has been exposed (eg, because of treatment or environmental exposure) to the investigational product prior to or around the time of conception and/or is exposed during his partner's pregnancy.

If a subject or subject's partner becomes or is found to be pregnant during the subject's treatment with the investigational product, the investigator must report this information to Pfizer Safety on the CT SAE Report Form and an EDP supplemental form, regardless of whether an SAE has occurred. In addition, the investigator must submit information regarding environmental exposure to a Pfizer product in a pregnant woman (eg, a subject reports that she is pregnant and has been exposed to a cytotoxic product by inhalation or spillage) to Pfizer Safety using the EDP supplemental form. This must be done irrespective of whether an AE has occurred and within 24 hours of awareness of the exposure. The information submitted should include the anticipated date of delivery (see below for information related to termination of pregnancy).

Follow-up is conducted to obtain general information on the pregnancy and its outcome for all EDP reports with an unknown outcome. The investigator will follow the pregnancy until completion (or until pregnancy termination) and notify Pfizer Safety of the outcome as a follow-up to the initial EDP supplemental form. In the case of a live birth, the structural integrity of the neonate can be assessed at the time of birth. In the event of a termination, the reason(s) for termination should be specified and, if clinically possible, the structural integrity of the terminated fetus should be assessed by gross visual inspection (unless preprocedure test findings are conclusive for a congenital anomaly and the findings are reported).

If the outcome of the pregnancy meets the criteria for an SAE (ie, ectopic pregnancy, spontaneous abortion, intrauterine fetal demise, neonatal death, or congenital anomaly [in a live-born baby, a terminated fetus, an intrauterine fetal demise, or a neonatal death]), the investigator should follow the procedures for reporting SAEs.

Additional information about pregnancy outcomes that are reported to Pfizer Safety as SAEs follows:

- Spontaneous abortion includes miscarriage and missed abortion;
- Neonatal deaths that occur within 1 month of birth should be reported, without regard to causality, as SAEs. In addition, infant deaths after 1 month should be reported as SAEs when the investigator assesses the infant death as related or possibly related to exposure to the investigational product.

Additional information regarding the EDP may be requested by the sponsor. Further follow-up of birth outcomes will be handled on a case-by-case basis (eg, follow-up on preterm infants to identify developmental delays). In the case of paternal exposure, the investigator will provide the subject with the Pregnant Partner Release of Information Form to deliver to his partner. The investigator must document in the source documents that the subject was given the Pregnant Partner Release of Information Form to provide to his partner.

# 8.4.3.2. Exposure During Breastfeeding

Scenarios of exposure during breastfeeding must be reported, irrespective of the presence of an associated SAE, to Pfizer Safety within 24 hours of the investigator's awareness, using the CT SAE Report Form. An exposure during breastfeeding report is not created when a Pfizer drug specifically approved for use in breastfeeding women (eg, vitamins) is administered in accord with authorized use. However, if the infant experiences an SAE associated with such a drug's administration, the SAE is reported together with the exposure during breastfeeding.

#### 8.4.3.3. Occupational Exposure

An occupational exposure occurs when, during the performance of job duties, a person (whether a healthcare professional or otherwise) gets in unplanned direct contact with the product, which may or may not lead to the occurrence of an AE.

An occupational exposure is reported to Pfizer Safety within 24 hours of the investigator's awareness, using the CT SAE Report Form, regardless of whether there is an associated SAE. Since the information does not pertain to a subject enrolled in the study, the information is not recorded on a CRF; however, a copy of the completed CT SAE Report Form is maintained in the investigator site file.

#### **8.4.4.** Medication Errors and Lack of Efficacy

Other exposures to the investigational product under study may occur in clinical trial settings, such as medication errors and lack of efficacy.

| Safety Event | Recorded on the CRF | Reported on the CT SAE<br>Report Form to Pfizer<br>Safety Within 24 Hours of |
|---|---|---|
| | | Awareness |
| Medication errors and lack of | All (regardless of whether | Only if associated with an |
| efficacy | associated with an AE) | SAE |

#### 8.4.4.1. Medication Errors

Medication errors may result from the administration or consumption of the investigational product by the wrong subject, or at the wrong time, or at the wrong dosage strength.

Medication errors include:

- Medication errors involving subject exposure to the investigational product;
- Potential medication errors or uses outside of what is foreseen in the protocol that do or do not involve the participating subject;
- The administration of expired investigational product;
- The administration of an incorrect investigational product;
- The administration of an incorrect dosage;
- The administration of investigational product that has undergone temperature excursion from the specified storage range, unless it is determined by the sponsor that the investigational product under question is acceptable for use.

Such medication errors occurring to a study participant are to be captured on the medication error page of the CRF, which is a specific version of the AE page.

In the event of a medication dosing error, the sponsor should be notified immediately.

Whether or not the medication error is accompanied by an AE, as determined by the investigator, the medication error is recorded on the medication error page of the CRF and, if applicable, any associated AE(s), serious and nonserious, are recorded on an AE page of the CRF.

Medication errors should be reported to Pfizer Safety within 24 hours on a CT SAE Report Form **only when associated with an SAE**.

#### 8.4.4.2. Lack of Efficacy

Lack of efficacy in an approved indication (approved Prevnar 13 indication in this age group) should be reported as an SAE to Pfizer Safety.

# 8.5. Medical Device Complaint Reporting Requirements

All medical device complaints, regardless of whether the medical device complaint is associated with an AE, will be recorded on the applicable pages within the CRF. This includes potential incidents or malfunctions associated with the use of a medical device product. An incident or malfunction is an event that might have led to death or serious deterioration in health, or if it occurred again might lead to death or serious deterioration in health.

Pfizer is to be notified of all medical device complaints within 24 hours of the investigator's awareness of the event.

#### 9. DATA ANALYSIS/STATISTICAL METHODS

Detailed methodology for summary and statistical analyses of the data collected in this study is outlined here and further detailed in a statistical analysis plan (SAP), which will be maintained by the sponsor. The SAP may modify what is outlined in the protocol where appropriate; however, any major modifications of the primary endpoint definitions or their analyses will also be reflected in a protocol amendment.

# 9.1. Sample Size Determination

The study size is not based on any formal statistical hypothesis test. Approximately 188 infants per vaccine group are planned to be randomized. No hypothesis tests between vaccine groups are planned; therefore, no power calculations for comparison of vaccine groups are included.

With 188 subjects per arm, the probabilities of observing at least 1 AE, local reaction, or systemic event where the true rate is 0.5%, 1%, and  $\geq$ 5% are presented in Table 5.

Table 5. Probability of Observing at Least 1 AE, Local Reaction, or Systemic Event by Assumed True Event Rates

| Sample Size | Assumed True Event Rate of at Least 1 AE, Local Reaction, or Systemic Event | | |
|---|---|---|---|
| | 0.5% | 1% | ≥5% |
| N = 188 | 0.610 | 0.849 | >0.999 |

# 9.2. Analysis Populations

The safety population will include all Group 1 and Group 2 subjects who receive at least 1 dose of c7vPnC and all Group 3 subjects who receive at least 1 dose of Prevnar 13. Subjects will be assigned to vaccine groups corresponding to the vaccine series actually received. The safety population will be the only analysis population for the primary endpoints.

The Dose 3 evaluable immunogenicity population will include any subject:

1. Who was eligible for the study.

- 2. Who was randomized and met the SAP-specified age window on the first day of vaccination for the randomized group (age windows will be same for Groups 1 and 3, but different for Group 2).
- 3. Who received c7vPnC and/or Prevnar 13, as randomly assigned, through Dose 3.
- 4. Who had an IgG concentration for at least 1 serotype 1 month after Dose 3.
- 5. Whose blood collection was within the SAP-specified window after Dose 3.
- 6. Who had no other major protocol deviations as determined by the clinician or medical monitor.

Additional criteria may be described in the SAP. The Dose 3 evaluable immunogenicity population will be the primary analysis population for immunogenicity results from the blood collected 1 month after Dose 3.



The Dose 4 evaluable immunogenicity population will include any subject:

- 1. Who was eligible for the study.
- 2. Who was randomized and met the SAP-specified age window on first day of vaccination for the randomized group (age windows will be same for Groups 1 and 3, but different for Group 2).
- 3. Who received the assigned vaccine, as randomized, within the defined window for Dose 4 as specified in the SAP.
- 4. Who received the vaccine to which he or she was randomly assigned at all 4 doses.
- 5. Who had an IgG concentration for at least 1 serotype 1 month after Dose 4.
- 6. Whose blood collection was within the SAP-specified window after Dose 4.
- 7. Who had no other major protocol deviations as determined by the clinician or medical monitor.

Additional criteria are described in the SAP. The Dose 4 evaluable immunogenicity population will be the primary analysis population for immunogenicity results after Dose 4.





# 9.3. Immunogenicity Analysis

All serotypes will be analyzed in the same way. All endpoints will be summarized by vaccine group.

9.3.1. Analyses of Secondary CCI Endpoints

The secondary CCl endpoints will be summarized by:

1. Geometric mean concentrations (GMCs) after Dose 3,

CCI

- 3. GMCs after Dose 4,
- 4. Proportions of subjects with IgG concentrations ≥ reference concentration after Dose 3,



Ninety-five percent confidence intervals (CIs) will also be calculated for all descriptive statistics.

GMCs and their CIs will be obtained by taking log transforms of concentrations, calculating the 95% CI with reference to the t-distribution, then exponentiating the mean and the limits. The Luminex assay IgG concentration of 0.35  $\mu$ g/mL will be used as the predefined IgG reference concentration for all serotypes, with the exception of serotypes 5 (0.23  $\mu$ g/mL), 6B (0.1  $\mu$ g/mL), and 19A (0.12  $\mu$ g/mL). The 95% CIs will be obtained using the Clopper-Pearson method.<sup>70</sup>





# 9.4. Safety Analysis

All safety analyses will be performed using the safety population.

Descriptive statistics for local reactions for the c7vPnC injection site in Groups 1 and 2 and the Supplemental Dose in Group 3, as well as the Prevnar 13 site in Group 3, and systemic events from Day 1 to Day 7 will be presented by severity and cumulatively across severity levels. Descriptive statistics will include proportions of subjects with the indicated endpoint and the associated Clopper-Pearson 95% CIs. Local reactions will be compiled for each dose for each group (Doses 1, 2, 3, and 4 and the Supplemental Dose) separately and compiled across all 4 doses of the same group.

AEs (including nonserious AEs, SAEs, and NDCMCs) will be compiled over 2 intervals: from Dose 1 to 1 month following Dose 3 and from Dose 4 to 1 month following Dose 4/Supplemental Dose. SAEs and NDCMCs will be summarized from Dose 1 until 6 months after Dose 4/Supplemental Dose. The descriptive statistics for AEs will be summarized as the number and percentage of subjects reporting at least 1 event of each preferred term with the associated Clopper-Pearson 95% CIs, arranged by system organ class.





# 10. QUALITY CONTROL AND QUALITY ASSURANCE

Pfizer or its agent will conduct periodic monitoring visits during study conduct to ensure that the protocol and GCPs are being followed. The monitors may review source documents to confirm that the data recorded on CRFs are accurate. The investigator and institution will allow Pfizer monitors/auditors or its agents and appropriate regulatory authorities direct access to source documents to perform this verification. This verification may also occur after study completion.

During study conduct and/or after study completion, the investigator site may be subject to review by the IRB/EC, and/or to quality assurance audits performed by Pfizer, or companies working with or on behalf of Pfizer, and/or to inspection by appropriate regulatory authorities.

The investigator(s) will notify Pfizer or its agents immediately of any regulatory inspection notification in relation to the study. Furthermore, the investigator will cooperate with Pfizer or its agents to prepare the investigator site for the inspection and will allow Pfizer or its agent, whenever feasible, to be present during the inspection. The investigator site and investigator will promptly resolve any discrepancies that are identified between the study data and the subject's medical records. The investigator will promptly provide copies of the inspection findings to Pfizer or its agent. Before response submission to the regulatory authorities, the investigator will provide Pfizer or its agents with an opportunity to review and comment on responses to any such findings.

It is important that the investigator(s) and their relevant personnel are available during the monitoring visits and possible audits or inspections and that sufficient time is devoted to the process.

#### 11. DATA HANDLING AND RECORD KEEPING

# 11.1. Case Report Forms/Electronic Data Record

As used in this protocol, the term CRF should be understood to refer to either a paper form or an electronic data record or both, depending on the data collection method used in this study.

A CRF is required and should be completed for each included subject. The completed original CRFs are the sole property of Pfizer and should not be made available in any form to third parties, except for authorized representatives of Pfizer or appropriate regulatory authorities, without written permission from Pfizer.

The investigator has ultimate responsibility for the collection and reporting of all clinical, safety, and laboratory data entered on the CRFs and any other data collection forms (source documents) and ensuring that they are accurate, authentic/original, attributable, complete, consistent, legible, timely (contemporaneous), enduring, and available when required. The CRFs must be signed by the investigator or by an authorized staff member to attest that the data contained on the CRFs are true. Any corrections to entries made in the CRFs or source documents must be dated, initialed, and explained (if necessary) and should not obscure the original entry.

In most cases, the source documents are the hospital or the physician subject chart. In these cases, data collected on the CRFs must match the data in those charts.

In some cases, the CRF may also serve as the source document. In these cases, a document should be available at the investigator site and at Pfizer that clearly identifies those data that will be recorded on the CRF, and for which the CRF will stand as the source document.

#### 11.2. Record Retention

To enable evaluations and/or inspections/audits from regulatory authorities or Pfizer, the investigator agrees to keep records, including the identity of all participating subjects (sufficient information to link records, eg, CRFs and hospital records), all original signed informed consent documents, copies of all CRFs, safety reporting forms, source documents, and detailed records of treatment disposition, and adequate documentation of relevant correspondence (eg, letters, meeting minutes, and telephone call reports). The records should be retained by the investigator according to the ICH guidelines, according to local regulations, or as specified in the clinical study agreement (CSA), whichever is longer.

If the investigator becomes unable for any reason to continue to retain study records for the required period (eg, retirement, relocation), Pfizer should be prospectively notified. The study records must be transferred to a designee acceptable to Pfizer, such as another investigator, another institution, or an independent third party arranged by Pfizer.

Investigator records must be kept for a minimum of 15 years after completion or discontinuation of the study or for longer if required by applicable local regulations.

The investigator must obtain Pfizer's written permission before disposing of any records, even if retention requirements have been met.

#### 12. ETHICS

#### 12.1. Institutional Review Board/Ethics Committee

It is the responsibility of the investigator to have prospective approval of the study protocol, protocol amendments, informed consent documents, and other relevant documents, eg, recruitment advertisements, if applicable, from the IRB/EC. All correspondence with the IRB/EC should be retained in the investigator file. Copies of IRB/EC approvals should be forwarded to Pfizer.

The only circumstance in which an amendment may be initiated prior to IRB/EC approval is where the change is necessary to eliminate apparent immediate hazards to the subjects. In that event, the investigator must notify the IRB/EC and Pfizer in writing immediately after the implementation.

# 12.2. Ethical Conduct of the Study

The study will be conducted in accordance with the protocol, legal and regulatory requirements, and the general principles set forth in the International Ethical Guidelines for Biomedical Research Involving Human Subjects (Council for International Organizations of Medical Sciences [CIOMS] 2002), ICH Guideline for Good Clinical Practice, and the Declaration of Helsinki.

# 12.3. Subject Information and Consent

All parties will ensure protection of subject personal data and will not include subject names or other identifiable data in any reports, publications, or other disclosures, except where required by law.

When study data are compiled for transfer to Pfizer and other authorized parties, subject names, addresses, and other identifiable data will be replaced by numerical codes based on a numbering system provided by Pfizer in order to de-identify study subjects. The investigator site will maintain a confidential list of subjects who participated in the study, linking each subject's numerical code to his or her actual identity. In case of data transfer, Pfizer will maintain high standards of confidentiality and protection of subjects' personal data consistent with applicable privacy laws.

The informed consent documents and any subject recruitment materials must be in compliance with ICH GCP, local regulatory requirements, and legal requirements, including applicable privacy laws.

The informed consent documents used during the informed consent process and any subject recruitment materials must be reviewed and approved by Pfizer, approved by the IRB/EC before use, and available for inspection.

The investigator must ensure that each study subject's legally acceptable representative is fully informed about the nature and objectives of the study and possible risks associated with participation.

Whenever consent is obtained from a subject's legally acceptable representative, the subject's assent (affirmative agreement) must subsequently be obtained when the subject has the capacity to provide assent, as determined by the IRB/EC. If the investigator determines that a subject's decisional capacity is so limited he/she cannot reasonably be consulted, then, as permitted by the IRB/EC and consistent with local regulatory and legal requirements, the subject's assent may be waived with source documentation of the reason assent was not obtained. If the study subject does not provide his or her own consent, the source documents must record why the subject did not provide consent (eg, minor, decisionally impaired adult), how the investigator determined that the person signing the consent was the subject's legally acceptable representative, the consent signer's relationship to the study subject (eg, parent, spouse), and that the subject's assent was obtained or waived. If assent is obtained verbally, it must be documented in the source documents.

The investigator, or a person designated by the investigator, will obtain written informed consent from each subject's legally acceptable representative before any study-specific activity is performed. The investigator will retain the original of each subject's signed consent document.

# 12.4. Reporting of Safety Issues and Serious Breaches of the Protocol or ICH GCP

In the event of any prohibition or restriction imposed (ie, clinical hold) by an applicable regulatory authority in any area of the world, or if the investigator is aware of any new

information that might influence the evaluation of the benefits and risks of the investigational product, Pfizer should be informed immediately.

In addition, the investigator will inform Pfizer immediately of any urgent safety measures taken by the investigator to protect the study subjects against any immediate hazard, and of any serious breaches of this protocol or of ICH GCP that the investigator becomes aware of.

#### 13. DEFINITION OF END OF TRIAL

# 13.1. End of Trial in All Participating Countries

End of trial in all participating countries is defined as last subject last visit (LSLV). After this time, sites will be closed out, the IRB/EC will be informed, and no further CIOMS reports will be sent.

#### 14. SPONSOR DISCONTINUATION CRITERIA

Premature termination of this study may occur because of a regulatory authority decision, change in opinion of the IRB/EC, or investigational product safety problems, or at the discretion of Pfizer. In addition, Pfizer retains the right to discontinue development of c7vPnC at any time.

If a study is prematurely terminated, Pfizer will promptly notify the investigator. After notification, the investigator must contact all participating subjects and the hospital pharmacy (if applicable) within 30 days. As directed by Pfizer, all study materials must be collected and all CRFs completed to the greatest extent possible.

#### 15. PUBLICATION OF STUDY RESULTS

# 15.1. Communication of Results by Pfizer

Pfizer fulfills its commitment to publicly disclose clinical trial results through posting the results of studies on www.clinicaltrials.gov (ClinicalTrials.gov), the European Clinical Trials Database (EudraCT), and/or www.pfizer.com, and other public registries in accordance with applicable local laws/regulations.

In all cases, study results are reported by Pfizer in an objective, accurate, balanced, and complete manner and are reported regardless of the outcome of the study or the country in which the study was conducted.

#### www.clinicaltrials.gov

Pfizer posts clinical trial US Basic Results on www.clinicaltrials.gov for Pfizer-sponsored interventional studies (conducted in patients) that evaluate the safety and/or efficacy of a Pfizer product, regardless of the geographical location in which the study is conducted. US Basic Results are submitted for posting within 1 year of the primary completion date (PCD) for studies in adult populations or within 6 months of the PCD for studies in pediatric populations.

Final Protocol Amendment 1, 18 Feb 2020

PCD is defined as the date that the final subject was examined or received an intervention for the purposes of final collection of data for the primary outcome, whether the clinical study concluded according to the prespecified protocol or was terminated.

#### **EudraCT**

Pfizer posts European Union (EU) Basic Results on EudraCT for all Pfizer-sponsored interventional studies that are in scope of EU requirements. EU Basic Results are submitted for posting within 1 year of the PCD for studies in adult populations or within 6 months of the PCD for studies in pediatric populations.

# www.pfizer.com

Pfizer posts Public Disclosure Synopses (clinical study report synopses in which any data that could be used to identify individual patients have been removed) on www.pfizer.com for Pfizer-sponsored interventional studies at the same time the US Basic Results document is posted to www.clinicaltrials.gov.

# 15.2. Publications by Investigators

Pfizer supports the exercise of academic freedom and has no objection to publication by the PI of the results of the study based on information collected or generated by the PI, whether or not the results are favorable to the Pfizer product. However, to ensure against inadvertent disclosure of confidential information or unprotected inventions, the investigator will provide Pfizer an opportunity to review any proposed publication or other type of disclosure of the results of the study (collectively, "publication") before it is submitted or otherwise disclosed.

The investigator will provide any publication to Pfizer at least 30 days before it is submitted for publication or otherwise disclosed. If any patent action is required to protect intellectual property rights, the investigator agrees to delay the disclosure for a period not to exceed an additional 60 days.

The investigator will, on request, remove any previously undisclosed confidential information before disclosure, except for any study- or Pfizer product-related information necessary to the appropriate scientific presentation or understanding of the study results.

If the study is part of a multicenter study, the investigator agrees that the first publication is to be a joint publication covering all investigator sites, and that any subsequent publications by the PI will reference that primary publication. However, if a joint manuscript has not been submitted for publication within 12 months of completion or termination of the study at all participating sites, the investigator is free to publish separately, subject to the other requirements of this section.

For all publications relating to the study, the institution will comply with recognized ethical standards concerning publications and authorship, including Section II - "Ethical Considerations in the Conduct and Reporting of Research" of the Uniform Requirements for

Manuscripts Submitted to Biomedical Journals, http://www.icmje.org/index.html#authorship, established by the International Committee of Medical Journal Editors.

Publication of study results is also provided for in the CSA between Pfizer and the institution. In this section entitled Publications by Investigators, the defined terms shall have the meanings given to them in the CSA.

If there is any conflict between the CSA and any attachments to it, the terms of the CSA control. If there is any conflict between this protocol and the CSA, this protocol will control as to any issue regarding treatment of study subjects, and the CSA will control as to all other issues.

#### 16. REFERENCES

- Said MA, Johnson HL, Nonyane BA, Deloria-Knoll M, O'Brien KL; for the AGEDD Adult Pneumococcal Burden Study Team. Estimating the burden of pneumococcal pneumonia among adults: a systematic review and meta-analysis of diagnostic techniques. *PLoS One*. 2013;8(4):e60273.
- O'Brien KL, Wolfson LJ, Watt JP, et al; for the Hib and Pneumococcal Global Burden of Disease Study Team. Burden of disease caused by *Streptococcus pneumoniae* in children younger than 5 years: global estimates. *Lancet*. 2009;374(9693):893-902.
- Huang SS, Johnson KM, Ray GT, et al. Healthcare utilization and cost of pneumococcal disease in the United States. *Vaccine*. 2011;29(18):3398-3412.
- Iyer AS, Ohtola JA, Westerink MAJ. Age-related immune response to pneumococcal polysaccharide vaccination: lessons for the clinic. *Expert Rev Vaccines*. 2015;14(1):85-97.
- Wahl B, O'Brien KL, Greenbaum A, et al. Global burden of *Streptococcus pneumoniae* in children younger than 5 years in the pneumococcal conjugate vaccines (PCV) era: 2000-2015. 10th International Symposium on Pneumococci & Pneumococcal Diseases (ISPPD-10); 26-30 Jun 2016; Glasgow, Scotland.
- <sup>6</sup> Centers for Disease Control and Prevention. Active Bacterial Core surveillance. Trends by serotype group, 1998-2015. http://www.cdc.gov/abcs/reportsfindings/survreports/spneu-types.html. Accessed 27 July 2016.
- Moore MR, Link-Gelles R, Schaffner W, et al. Effect of use of 13-valent pneumococcal conjugate vaccine in children on invasive pneumococcal disease in children and adults in the USA: analysis of multisite, population-based surveillance. *Lancet Infect Dis*. 2015;15(3):301-309.
- Olarte L, Barson WJ, Barson RM, et al. Impact of the 13-valent pneumococcal conjugate vaccine on pneumococcal meningitis in US children. *Clin Infect Dis*. 2015;61(5):767-775.
- Stockmann C, Ampofo K, Byington CL, et al. Pneumococcal meningitis in children: epidemiology, serotypes, and outcomes from 1997-2010 in Utah. *Pediatrics*. 2013;132(3):421-428.
- Jain S, Williams DJ, Arnold SR, et al; for the CDC EPIC Study Team. Community-acquired pneumonia requiring hospitalization among U.S. children. *N Engl J Med*. 2015;372(9):835-845.

- Jain S, Self WH, Wunderink RG, et al; for the CDC EPIC Study Team. Community-acquired pneumonia requiring hospitalization among U.S. adults. *N Engl J Med*. 2015;373(5):415-427.
- Marom T, Tan A, Wilkinson GS, Pierson K, Freeman JL, Chonmaitree T. Trends in otitis media–related health care use in the United States, 2001-2011. *JAMA Pediatr*. 2014;168(1):68-75.
- Geno KA, Gilbert GL, Song JY, et al. Pneumococcal capsules and their types: past, present, and future. *Clin Microbiol Rev.* 2015;28(3):871-899.
- Hausdorff WP, Hanage WP. Interim results of an ecological experiment—conjugate vaccination against the pneumococcus and serotype replacement. *Hum Vaccin Immunother*. 2016;12(2):358-374.
- AlonsoDeVelasco E, Verheul AFM, Verhoef J, Snippe H. *Streptococcus pneumoniae*: virulence factors, pathogenesis, and vaccines. *Microbiol Rev.* 1995;59(4):591-603.
- Prevention of pneumococcal disease: recommendations of the Advisory Committee on Immunization Practices (ACIP). *MMWR Recomm Rep.* 1997;46(RR-8):1-24.
- Austrian R. A brief history of pneumococcal vaccines. *Drugs Aging*. 1999;15(suppl 1):1-10.
- Shapiro ED, Berg AT, Austrian R, et al. The protective efficacy of polyvalent pneumococcal polysaccharide vaccine. *N Engl J Med.* 1991;325(21):1453-1460.
- Stein KE. Thymus-independent and thymus-dependent responses to polysaccharide antigens. *J Infect Dis.* 1992;165 suppl 1:S49-S52.
- Borrow R, Health PT, Siegrist CA. Use of pneumococcal polysaccharide vaccine in children: what is the evidence? *Curr Opin Infect Dis.* 2012;25(3):292-303.
- Jackson LA, Neuzil KM, Yu O, et al; for the Vaccine Safety Datalink. Effectiveness of pneumococcal polysaccharide vaccine in older adults. N Engl J Med. 2003;348(18):1747-1755.
- Leventer-Roberts M, Feldman BS, Brufman I, Cohen-Stavi CJ, Hoshen M, Balicer RD. Effectiveness of 23-valent pneumococcal polysaccharide vaccine against invasive disease and hospital-treated pneumonia among people aged ≥65 years: a retrospective case-control study. *Clin Infect Dis.* 2015;60(10):1472-1480.
- Wright PF, Sell SH, Vaughn WK, Andrews C, McConnell KB, Schiffman G. Clinical studies of pneumococcal vaccines in infants. II. Efficacy and effect on nasopharyngeal carriage. *Rev Infect Dis.* 1981;3 suppl:S108-S112.

- Torres A, Bonanni P, Hryniewicz W, Moutschen M, Reinert RR, Welte T. Pneumococcal vaccination: what have we learnt so far and what can we expect in the future? *Eur J Clin Microbiol Infect Dis*. 2015;34(1):19-31.
- Robinson KA, Baughman W, Rothrock G, et al; for the Active Bacterial Core Surveillance (ABCs)/Emerging Infections Program Network. Epidemiology of invasive *Streptococcus pneumoniae* infections in the United States, 1995-1998: opportunities for prevention in the conjugate vaccine era. *JAMA*. 2001;285(13):1729-1735.
- Hausdorff WP, Bryant J, Paradiso PR, Siber GR. Which pneumococcal serogroups cause the most invasive disease: implications for conjugate vaccine formulation and use, part I. *Clin Infect Dis*. 2000;30(1):100-121.
- Hausdorff WP, Bryant J, Kloek C, Paradiso PR, Siber GR. The contribution of specific pneumococcal serogroups to different disease manifestations: implications for conjugate vaccine formulation and use, part II. *Clin Infect Dis.* 2000;30(1):122-140.
- Nuorti JP, Whitney CG. Prevention of pneumococcal disease among infants and children use of 13-valent pneumococcal conjugate vaccine and 23-valent pneumococcal polysaccharide vaccine recommendations of the Advisory Committee on Immunization Practices (ACIP). *MMWR Recomm Rep.* 2010;59(RR-11):1-18.
- Johnson HL, Deloria-Knoll M, Levine OS, et al. Systematic evaluation of serotypes causing invasive pneumococcal disease among children under five: the Pneumococcal Global Serotype Project. *PLoS Med.* 2010;7(10):1-13.
- Richter SS, Heilmann KP, Dohrn CL, Riahi F, Diekema DJ, Doern GV. Pneumococcal serotypes before and after introduction of conjugate vaccines, United States, 1999-2011. *Emerg Infect Dis.* 2013;19(7):1074-1083.
- Black SB, Shinefield HR, Ling S, et al. Effectiveness of heptavalent pneumococcal conjugate vaccine in children younger than five years of age for prevention of pneumonia. *Pediatr Infect Dis J.* 2002;21(9):810-815.
- Hansen J, Black S, Shinefield H, et al. Effectiveness of heptavalent pneumococcal conjugate vaccine in children younger than 5 years of age for prevention of pneumonia: updated analysis using World Health Organization standardized interpretation of chest radiographs. *Pediatr Infect Dis J.* 2006;25(9):779-781.
- Cutts FT, Zaman SM, Enwere G, et al; for the Gambian Pneumococcal Vaccine Trial Group. Efficacy of nine-valent pneumococcal conjugate vaccine against pneumonia and invasive pneumococcal disease in The Gambia: randomised, double-blind, placebo-controlled trial. *Lancet*. 2005;365(9465):1139-1146.

- Eskola J, Kilpi T, Palmu A, et al; for the Finnish Otitis Media Study Group. Efficacy of a pneumococcal conjugate vaccine against acute otitis media. *N Engl J Med*. 2001;344(6):403-409.
- O'Brien KL, Moulton LH, Reid R, et al. Efficacy and safety of seven-valent conjugate pneumococcal vaccine in American Indian children: group randomised trial. *Lancet*. 2003;362(9381):355-361.
- Klugman KP, Madhi SA, Huebner RE, Kohberger R, Mbelle N, Pierce N; for the Vaccine Trialists Group. A trial of a 9-valent pneumococcal conjugate vaccine in children with and those without HIV infection. *N Engl J Med.* 2003;349(14):1341-1348.
- Pilishvili T, Lexau C, Farley MM, et al; for the Active Bacterial Core Surveillance/Emerging Infections Program Network. Sustained reductions in invasive pneumococcal disease in the era of conjugate vaccine. *J Infect Dis.* 2010;201(1):32-41.
- Reinert RR, Paradiso P, Fritzell B. Advances in pneumococcal vaccines: the 13-valent pneumococcal conjugate vaccine received market authorization in Europe. *Expert Rev Vaccines*. 2010;9(3):229-236.
- Bonten MJM, Huijts SM, Bolkenbaas M, et al. Polysaccharide conjugate vaccine against pneumococcal pneumonia in adults. *N Engl J Med*. 2015;372(12):1114-1125.
- Centers for Disease Control and Prevention. Licensure of a 13-valent pneumococcal conjugate vaccine (PCV13) and recommendations for use among children -- Advisory Committee on Immunization Practices (ACIP), 2010. *MMWR Morb Mortal Wkly Rep.* 2010;59(9):258-261.
- Centers for Disease Control and Prevention. Licensure of 13-valent pneumococcal conjugate vaccine for adults aged 50 years and older. *MMWR Morb Mortal Wkly Rep.* 2012;61(21):394-395.
- Prevenar 13 Summary of Product Characteristics.

  http://www.ema.europa.eu/docs/en\_GB/document\_library/EPAR\_\_Product\_Information/human/001104/WC500057247.pdf. Accessed 12 Sep 2016.
- European Medicines Agency. Prevenar 13 Assessment Report. 22 Jan 2015. http://www.ema.europa.eu/docs/en\_GB/document\_library/EPAR\_-\_Assessment\_Report\_-\_Variation/human/001104/WC500186805.pdf. Accessed 12 Sep 2016.
- World Health Organization. WHO Prequalified Vaccines. Pneumococcal (conjugate). Prevenar 13. https://extranet.who.int/gavi/PQ\_Web/PreviewVaccine.aspx?nav=0&ID=221. Effective 20 Aug 2010. Accessed 12 Sep 2016.

- World Health Organization. WHO Prequalified Vaccines. Pneumococcal (conjugate). Prevenar 13 Multidose Vial. https://extranet.who.int/gavi/PQ\_Web/PreviewVaccine.aspx?nav=0&ID=317. Effective 14 Jul 2016. Accessed 12 Sep 2016.
- Harboe ZB, Dalby T, Weinberger DM, et al. Impact of 13-valent pneumococcal conjugate vaccination in invasive pneumococcal disease incidence and mortality [erratum appears in *Clin Infect Dis*. 2014;59(12):1812]. *Clin Infect Dis*. 2014;59(8):1066-1073.
- Steens A, Bergsaker MA, Aaberge IS, Rønninga K, Vestrheimaa DF. Prompt effect of replacing the 7-valent pneumococcal conjugate vaccine with the 13-valent vaccine on the epidemiology of invasive pneumococcal disease in Norway. *Vaccine*. 2013;31(52):6232-6238.
- Miller E, Andrews NJ, Waight PA, Slack MPE, George RC. Effectiveness of the new serotypes in the 13-valent pneumococcal conjugate vaccine. *Vaccine*. 2011;29(49):9127-9131.
- Cohen R, Biscardi S, Levy C. The multifaceted impact of pneumococcal conjugate vaccine implementation in children in France between 2001 to 2014. *Hum Vaccines Immunother*. 2016;12(2):277-284.
- Cohen R, Levy C, Bingen E, Koskas M, Nave I, Varon E. Impact of 13-valent pneumococcal conjugate vaccine on pneumococcal nasopharyngeal carriage in children with acute otitis media. *Pediatr Infect Dis J.* 2012;31(3):297-301.
- Flasche S, Van Hoek AJ, Sheasby E, et al. Effect of pneumococcal conjugate vaccination on serotype-specific carriage and invasive disease in England: a cross-sectional study. *PLoS Med.* 2011;8(4):e1001017.
- Williams SR, Mernagh PJ, Lee MHT, Tan JT. Changing epidemiology of invasive pneumococcal disease in Australian children after introduction of a 7-valent pneumococcal conjugate vaccine. *Med J Aust*. 2011;194(3):116-120.
- Lepoutre A, Varon E, Georges S, Gutmann L, Lévy-Bruhl D. Impact of infant pneumococcal vaccination on invasive pneumococcal diseases in France, 2001-2006. *Euro Surveill*. 2008;13(35):18962.
- Munoz-Almagro C, Ciruela P, Esteva C, et al; for the Catalan Study Group of Invasive Pneumococcal Disease. Serotypes and clones causing invasive pneumococcal disease before the use of new conjugate vaccines in Catalonia, Spain. *J Infect*. 2011;63(2):151-162.

- Norton NB, Stanek RJ, Mufson MA. Routine pneumococcal vaccination of children provokes new patterns of serotypes causing invasive pneumococcal disease in adults and children. *Am J Med Sci.* 2013;345(2):112-120.
- Adam HJ, Karlowsky JA, Nichol KA, et al. Baseline epidemiology of *Streptococcus pneumoniae* serotypes in Canada prior to the introduction of the 13-valent pneumococcal vaccine. *Microb Drug Resist*. 2012;18(2):176-182.
- Gonzalez BE, Hulten KG, Lamberth L, Kaplan SL, Mason EO Jr; and the U.S. Pediatric Multicenter Pneumococcal Surveillance Group. *Streptococcus pneumoniae* serogroups 15 and 33: an increasing cause of pneumococcal infections in children in the United States after the introduction of the pneumococcal 7-valent conjugate vaccine. *Pediatr Infect Dis J.* 2006;25(4):301-305.
- Harboe ZB, Thomsen RW, Riis A, et al. Pneumococcal serotypes and mortality following invasive pneumococcal disease: a population-based cohort study. *PLoS Med*. 2009;6(5):e1000081.
- Wroe PC, Lee GM, Finkelstein JA, et al. Pneumococcal carriage and antibiotic resistance in young children before 13-valent conjugate vaccine. *Pediatr Infect Dis J.* 2012;31(3):249-254.
- Cohen R, Varon E, Doit C, et al. A 13-year survey of pneumococcal nasopharyngeal carriage in children with acute otitis media following PCV7 and PCV13 implementation. *Vaccine*. 2015;33(39):5118-5126.
- Demczuk WHB, Martin I, Griffith A, et al; Toronto Bacterial Diseases Network; Canadian Public Health Laboratory Network. Serotype distribution of invasive *Streptococcus pneumoniae* in Canada after the introduction of the 13-valent pneumococcal conjugate vaccine, 2010–2012. *Can J Microbiol*. 2013;59(12):778-788.
- <sup>62</sup> Cohen R, Cohen JF, Chalumeau M, Levy C. Impact of pneumococcal conjugate vaccines for children in high- and non-high-income countries. *Expert Rev Vaccines*. 2017;16(6):625-640.
- Balsells E, Guillot L, Nair H, et al. Serotype distribution of *Streptococcus pneumoniae* causing invasive disease in children in the post-PCV era: a systematic review and meta-analysis. *PloS One*. 2017;12(5):e0177113.
- Golden AR, Adam HJ, Zhanel GG; Canadian Antimicrobial Resistance Alliance (CARA). Invasive *Streptococcus pneumoniae* in Canada, 2011–2014: characterization of new candidate 15-valent pneumococcal conjugate vaccine serotypes 22F and 33F. *Vaccine*. 2016;34(23):2527-2530.

- Metcalf BJ, Gertz RE Jr, Gladstone RA, et al. Strain features and distributions in pneumococci from children with invasive disease before and after 13-valent conjugate vaccine implementation in the USA. *Clin Microbiol Infect*. 2016;22(1):60.e9-.e29.
- Waight PA, Andrews NJ, Ladhani SN, Sheppard CL, Slack MPE, Miller E. Effect of the 13-valent pneumococcal conjugate vaccine on invasive pneumococcal disease in England and Wales 4 years after its introduction: an observational cohort study. *Lancet Infect Dis.* 2015;15(5):535-543.
- van der Linden M, Falkenhorst G, Perniciaro S, Imohl M. Effects of infant pneumococcal conjugate vaccination on serotype distribution in invasive pneumococcal disease among children and adults in Germany. *PLoS One*. 2015;10(7):e0131494.
- Prevnar 13 [package insert on FDA Website]. Philadelphia, PA: Wyeth Pharmaceuticals, Inc; 2016. https://www.fda.gov/downloads/BiologicsBloodVaccines/Vaccines/ApprovedProducts/UCM201669.pdf. Accessed 11 Dec 2017.
- <sup>69</sup> Food and Drug Administration, Center for Biologics Evaluation and Research. Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials. Guidance for Industry, September 2007.
- Collett D. *Modelling Binary Data*. London: Chapman & Hall; 1991.

# **Appendix 1. Abbreviations**

The following is a list of abbreviations that may be used in the protocol.

| Abbreviation | Term |
|--------------|-------------------------------------------------------------|
| AE | adverse event |
| ALT | alanine aminotransferase |
| AOM | acute otitis media |
| AST | aspartate aminotransferase |
| c7vPnC | complementary 7-valent pneumococcal conjugate vaccine |
| CAP | community-acquired pneumonia |
| CBER | Center for Biologics Evaluation and Research |
| CDC | Centers for Disease Control and Prevention |
| CI | confidence interval |
| CIOMS | Council for International Organizations of Medical Sciences |
| CK | creatine kinase |
| CRF | case report form |
| CRM197 | cross-reactive material 197 |
| CSA | clinical study agreement |
| CT | clinical trial |
| DILI | drug-induced liver injury |
| DTaP | diphtheria, tetanus, and acellular pertussis |
| EC | ethics committee |
| e-diary | electronic diary |
| CCI | |
| ELISA | enzyme-linked immunosorbent assay |
| EU | European Union |
| EudraCT | European Clinical Trials Database |
| FDA | Food and Drug Administration |
| GCP | Good Clinical Practice |
| GGT | gamma-glutamyl transferase |
| GMC | geometric mean concentration |
| CCI | |
| GMT | geometric mean titer |
| IB | investigator's brochure |
| ICH | International Council for Harmonisation |
| ID | identification |
| IgG | immunoglobulin G |
| IM | intramuscularly |
| IND | investigational new drug application |
| INR | international normalized ratio |
| IP | investigational product |
| IPD | invasive pneumococcal disease |
| IRB | institutional review board |
| CCI | |
| IRT | interactive response technology |
| IU | international units |

| Abbreviation | Term |
|--------------|-----------------------------------------------|
| IWR | interactive Web-based response |
| LFT | liver function test |
| LLOQ | lower limit of quantitation |
| LSLV | last subject last visit |
| MMR | measles, mumps, and rubella |
| N/A | not applicable |
| NDCMC | newly diagnosed chronic medical condition |
| OPA | opsonophagocytic activity |
| PCD | primary completion date |
| PI | principal investigator |
| PPSV23 | 23-valent pneumococcal polysaccharide vaccine |
| PT | prothrombin time |
| CCI | |
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| SRM | study reference manual |
| SRSD | single reference safety document |
| TBili | total bilirubin |
| ULN | upper limit of normal |
| US | United States |
| USPI | US package insert |
| VT | vaccine-type |
| WHO | World Health Organization |

# **Document Approval Record**

| Document Name: | C3571002 Protocol Amendment 1 Clean Copy 18Feb2020 |
|----------------|----------------------------------------------------|
|----------------|----------------------------------------------------|

Document Title:

A PHASE 2, RANDOMIZED, OPEN-LABEL TRIAL TO EVALUATE THE SAFETY AND IMMUNOGENICITY OF A MULTIVALENT PNEUMO COCCAL CONJUGATE VACCINE GIVEN WITH, OR SEPARATELY FROM, 13-VALENT PNEUMOCOCCAL CONJUGATE VACCINE IN HE

**ALTHY INFANTS** 

| Signed By: | Date(GMT) | Signing Capacity |
|------------|----------------------|------------------|
| PPD | 20-Feb-2020 21:47:45 | Final Approval |
| PPD | 21-Feb-2020 18:19:06 | Final Approval |